A Double-Blind, Randomized, Parallel-Group Study to Evaluate the Efficacy, Safety and Tolerability of Fixed Dose Combination GSP 301 Nasal Spray Compared With Placebo Nasal Spray in Pediatric Subjects (Aged 6 to Under 12 Years) With Seasonal Allergic Rhinitis (SAR)

Identifiers

NCT03463031

Date of Document

06 December 2018

# STATISTICAL ANALYSIS PLAN PHASE III

VERSION: FINAL DATE OF PLAN:

06-DEC-2018

#### **BASED ON:**

GSP 301-305 Protocol Version 3.0, 18-July-2018

#### **STUDY DRUG:**

Fixed Dose Combination of Olopatadine Hydrochloride and Mometasone Furoate, GSP 301 Nasal Spray (NS)

#### PROTOCOL NUMBER:

GSP 301-305

# STUDY TITLE:

A Double-Blind, Randomized, Parallel-Group Study to Evaluate the Efficacy, Safety and Tolerability of Fixed Dose Combination GSP 301 Nasal Spray Compared with Placebo Nasal Spray in Pediatric Subjects (Aged 6 to Under 12 Years) with Seasonal Allergic Rhinitis (SAR)

#### **SPONSOR:**

Glenmark Specialty S.A. Avenue Léopold-Robert 37 2300 La Chaux-de-Fonds Switzerland

This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

# SIGNATURE PAGE

This document has been prepared and reviewed by:

Senior Statistician Chiltern Senior I appri 06 De

Senior Biostatistician 1 I approved this document 06 Dec 2018 10:35 PM -05:00

Signature

Date

This document has been reviewed and approved by:

Senior Principal Statistician Clinical Operations-Biometrics Glenmark Specialty S.A.



OFFECZOR

# **TECHNICAL SUMMARY REPORT (TSR)**

#### Name of Sponsor/Company:

Glenmark Specialty S.A.

Name of Study Drug: GSP 301 NS - Fixed dose combination of olopatadine hydrochloride and mometasone furoate

#### Title of Study:

A Double-Blind, Randomized, Parallel-Group Study to Evaluate the Efficacy, Safety and Tolerability of Fixed Dose Combination GSP 301 Nasal Spray Compared with Placebo Nasal Spray in Pediatric Subjects (Aged 6 to Under 12 Years) with Seasonal Allergic Rhinitis (SAR)

IND no: 123164 EudraCT no: Not applicable

Indication: Seasonal allergic rhinitis (SAR)

#### Investigators:

Study Center(s): Approximately 40 sites in the United States

#### Studied period:

Subject participation may be 22 days up to 27 days with 7 to 10 days of a screening/run-in period and a 14-day treatment period, with allowable window periods for the study visits.

Phase of development: Phase III

#### **Objectives:**

#### Primary:

To compare the efficacy of GSP 301 Nasal Spray (NS) with GSP 301 placebo NS over 14 days of study treatment in pediatric subjects (aged  $\geq$ 6 to <12 years) with SAR.

#### Secondary:

To assess the safety and tolerability of each treatment over 14 days of study treatment in pediatric subjects (aged >6 to <12 years) with SAR.

**Study population:** Male and non-pregnant female subjects aged ≥6 to <12 years with documented clinical history of SAR (for at least 2 years preceding the Screening Visit) with exacerbations (clinical evidence of active symptoms) during the spring or fall allergy seasons for the relevant seasonal allergen (eg, tree/grass pollen or ragweed pollen).

Study design/ Methodology: This is a phase 3, double-blind, randomized, parallel-group, placebo-controlled, multicenter study to compare the efficacy and safety of GSP 301 NS with placebo NS in pediatric subjects (aged ≥6 to <12 years) with SAR. The subject participation may be 22 days up to 27 days with 7 to 10 days of a screening/placebo run-in period and 14 days of treatment period, with allowable window periods for the study visits. Enrollment will complete when subjects have been randomized to treatment.

December 06, 2018

# Number of Subjects (planned and analyzed):

A total of approximately 450 subjects (225 subjects per treatment group) are planned to be randomized to treatment during this study.

#### Diagnosis and main criteria for inclusion (see protocol section 7):

The subject population will be Pediatric Subjects (Aged 6 to Under 12 Years) who exhibit symptoms of SAR during the spring or fall allergy season, as applicable.

#### Inclusion Criteria

Subjects eligible for enrolment in the study must meet all of the following criteria:

- 1. Male or non-pregnant female subjects aged ≥6 to <12 years, at the Screening Visit (Visit 1).
- 2. Signed informed consent/assent form (subject and parent/caregiver/legal guardian), which meets all criteria of the current Food and Drug Administration/local regulations.
- 3. Documented clinical history of SAR (for at least 2 years preceding the Screening Visit [Visit 1]) with exacerbations (clinical evidence of active symptoms) during the study season for the relevant seasonal allergen (eg, tree/grass pollen or ragweed pollen). SAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past, and in the Investigator's judgment, is expected to require treatment throughout the study period.
- 4. Demonstrated sensitivity to at least 1 seasonal allergen (eg, tree/grass pollen or ragweed pollen) known to induce SAR through a documented positive skin prick test (wheal diameter at least 5 mm greater than the negative control) to a relevant seasonal allergen. Documentation of a positive result within 12 months prior to the Screening Visit (Visit 1) is acceptable. The subject's positive allergen must be consistent with the medical history of SAR. Additionally, the subject is expected to be adequately exposed to the SAR allergen that he/she has tested positive for the entire duration of the study.
- 5. A 12-hour reflective Total Nasal Symptom Score (rTNSS) value of ≥6 (out of a possible 12) for the morning (AM) assessment at the Screening Visit (Visit 1).
- 6. General good health and free of any disease or concomitant treatment that could interfere with the interpretation of study results, as determined by the Investigator.
- 7. Able to demonstrate the correct NS application technique (with the help of parents/guardians/caregivers, if needed) at the Screening Visit (Visit 1).
- 8. Willing and able to comply with all aspects of the protocol (with the help of parents/guardians/caregivers, if needed).

#### Exclusion Criteria

Subjects meeting any of the following criteria must not be enrolled in the study:

- 1. Eligible females of childbearing potential who are known to be sexually active or pregnant, will be excluded and referred for appropriate evaluation. If a girl has reached puberty and achieved menarche (as determined by the Investigator), parents/guardians/caregivers will be consulted to obtain consent for pregnancy testing and permission to counsel the subject followed by counselling the subject by the Investigator regarding the possible unknown risks associated with study medication during pregnancy. Urine pregnancy test must be negative at the Screening Visit (Visit 1). Male subjects who are known to be sexually active will also be excluded and referred appropriately.
- 2. Plans to travel outside the known pollen area for the investigational site for 24 hours or longer during the last 7 days of the screening/run-in period.
- 3. Plans to travel outside the known pollen area for the investigational site for 2 or more consecutive days OR 3 or more days in total between the Randomization Visit (Visit 2) and the Final Treatment Visit (Visit 4).

- 4. History of significant (based on Investigator's judgement) atopic dermatitis or rhinitis medicamentosa (within 60 days prior to the Screening Visit [Visit 1])
- 5. Treatment with any known strong cytochrome P450 (CYP)3A4 inducers (eg, carbamazepine, phenytoin, rifabutin, rifampin, pioglitazone etc.) or strong inhibitors (eg, azole antifungals, macrolide antibiotics) within 30 days prior to the Screening Visit (Visit 1), or during the study.
- 6. Non-vaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding Screening Visit (Visit 1).
- 7. A known hypersensitivity to any corticosteroids or antihistamines or to either of the drug components of the Investigational Product or its excipients.
- 8. History of anaphylaxis and/or other severe local reaction(s) to skin testing.
- 9. Any history or current use of alcohol or drug dependence at the Screening Visit (Visit 1), as determined by the Investigator.
- 10. History of positive test for human immunodeficiency virus, Hepatitis B or Hepatitis C infection (parents/guardians/caregivers will be consulted to obtain consent).
- 11. History and evidence of acute or significant chronic sinusitis or chronic purulent post nasal drip at the Screening Visit (Visit 1).
- 12. Any of the following conditions (including but not limited to the following) that are judged by the Investigator to be clinically significant and/or to affect the subject's ability to participate in this study:
  - impaired hepatic function.
  - any systemic infection.
  - hematological, hepatic, renal, endocrine disorder (except for hypothyroidism).
  - gastrointestinal disease.
  - malignancy (excluding basal cell carcinoma).
  - current neuropsychological condition with or without drug therapy.
    - Subjects with history or current diagnosis of active Attention Deficit Hyperactivity Disorder (ADHD) can be included in the study if symptoms of ADHD are considered stable by the treating physician and such history is documented by the Investigator.
    - Subjects with history or current diagnosis of ADHD on medications are eligible for inclusion if they are on stable active drug therapy and have stable symptoms for at least 30 days before the screening visit as documented in the medical history by the Investigator. Subjects may not be withdrawn from ADHD treatment medications during screening and/or throughout the study. If ADHD treatment medications are planned to be withdrawn or withdrawn by the treating physician during the study, then the subject should be considered ineligible or early terminated, respectively.
  - cardiovascular disease (eg, uncontrolled hypertension).
  - respiratory disease other than mild asthma.
- 13. Any major surgery (as assessed by the Investigator) within 4 weeks before the Screening Visit (Visit 1).
- 14. A requirement for the chronic use of tricyclic anti-depressants.
- 15. Dependence (in the opinion of the Investigator) on nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids.
- 16. Active pulmonary disorder or infection (including but not limited to bronchitis, pneumonia, or influenza), upper respiratory tract or sinus infection within the 14 days prior to the Screening Visit (Visit 1) or the development of respiratory infections during the placebo run-in period. Subjects with mild asthma (as

- judged by the Investigator) are allowable on the condition that treatment is limited to inhaled short-acting beta agonists only (up to 8 puffs per day).
- 17. Use of antibiotic therapy for acute conditions within 14 days prior to Screening Visit (Visit 1). Low doses of antibiotics taken for prophylaxis are allowed if the therapy was started prior to the Screening Visit (Visit 1) and is expected to continue at the same stable dose throughout the clinical study duration.
- 18. Posterior subcapsular cataracts or glaucoma, or any other ocular disturbances or other listed related conditions (as applicable) including:
  - · history of increased intraocular pressure.
  - history of retinal detachment surgery.
  - history of incisional eye surgery (other than unilateral cataract extraction or laser-assisted in situ keratomileusis).
  - history of penetrating ocular trauma, severe blunt ocular trauma.
  - evidence of uveitis, iritis, or other inflammatory eye disease during screening.
  - presence of ocular herpes simplex.
- 19. Known history of hypothalamic-pituitary-adrenal axis impairment.
- 20. Existence of any significant surgical or medical condition, or clinically significant physical finding (eg, significant nasal polyps or other clinically significant respiratory tract malformations/nasal structural abnormalities, significant nasal trauma [such as nasal piercing] or significant nasal septal deviation) which, in the opinion of the Investigator (or in consultation with the Sponsor's medical monitor/designee), significantly interferes with the absorption, distribution, metabolism or excretion of the study medication or significantly interferes with nasal air flow or interferes with the subject's ability to reliably complete the AR Assessment Diary.
- 21. Participation in any investigational non-biological drug clinical study in the 30 days or investigational biological drug in the 120 days preceding the Screening Visit (Visit 1) or planned participation in another investigational clinical study at any time during the current study.
- 22. Initiation of immunotherapy injections or immunosuppressive/immune-modulator medications within 60 days preceding the Screening Visit (Visit 1) and/or currently undergoing treatment with immunotherapy or immunosuppressive/immune-modulator medications. Topical pimecrolimus cream or tacrolimus ointment treatment if initiated at least 30 days prior to screening and maintained on stable dose is acceptable. A 180-day washout period is required following the last dose of sublingual immunotherapy (investigational or other) prior to the Screening Visit (Visit 1).
- 23. Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone, or equivalent, within 30 days prior to the Screening Visit (Visit 1); use of a topical hydrocortisone or equivalent in any concentration covering greater than 20% of the body surface or the presence of an underlying condition (as judged by the Investigator) that can reasonably be expected to require treatment with such preparations over the clinical study duration.
- 24. Previous participation in another GSP 301 NS study as a randomized subject.
- 25. Clinical study participation by clinical investigator site employees and/or their immediate relatives.
- 26. Study participation by more than 1 subject from the same household at the same time. However, after the completion/discontinuation by 1 subject in the household, another subject from the same household may be screened.
- 27. Known to have failed to show symptom improvement with any approved/marketed monotherapy component of the GSP 301 NS (ie, NASONEX NS, PATANASE NS, or both) as judged by the Investigator.

Randomization Criteria (at the Randomization Visit (RV) – Visit 2)

- 1. Continued general good health and continued eligibility according to the inclusion and exclusion criteria.
- 2. Has not left the known pollen area for the investigative site for 24 hours or longer during the last 7 days of the placebo run-in period.
- 3. No adverse event (AE) that has altered eligibility according to the inclusion and exclusion criteria.
- 4. Minimum 12-hour subject-reported rTNSS of an average of 6, (out of a possible 12) during the last 4 days of the placebo run-in period (average of last 8 consecutive AM and PM assessments from the Day -4 PM assessment to the AM assessment on the day of randomization).
- 5. A 12-hour subject-reported reflective nasal congestion score of an average of 2 or greater during the last 4 days of the placebo run-in period (average of last 8 consecutive AM and PM assessments from Day -4 PM assessment to the AM assessment on the day of randomization).
- 6. Adequate symptom assessment diary compliance (with assistance from parent/guardian/caregiver, as needed) inadequate compliance is defined as missing one or more of the entries on 2 or more assessment sessions (AM or PM) during the last 4 days of the placebo run-in period (during the last 8 consecutive AM and PM assessments from Day -4 PM assessment to the AM assessment on the day of randomization).
- 7. Adequate study medication compliance each subject must have taken his/her single-blind placebo medication (with assistance from parent/guardian/caregiver, as needed) for at least 80% of the entire placebo run-in period as reported in the symptom assessment diary.
- 8. Absence of common cold, upper respiratory infections, otitis, lower respiratory infections or acute sinusitis for 14 days prior to the Randomization Visit (Visit 2).
- 9. No use of prohibited concomitant medications during the placebo run-in period.

#### Study-Specific Discontinuation/Withdrawal Criteria:

A subject (or parent/guardian, as applicable) may voluntarily discontinue study participation at any time after giving informed consent/assent and before the completion of the last visit of the study. Subjects may also be withdrawn from study drug treatment at the discretion of the Investigator or Sponsor for safety, noncompliance, or administrative reasons. The Investigator may also discontinue the subject's study participation at any time at his/her discretion and for any reason.

The reasons for subject withdrawal will be recorded and may include, but are not limited to:

- 1. Withdrawal of consent/assent by the subject (or parent/legal guardian, as applicable) to continue in the study. If consent is withdrawn, the subject will not receive any further investigational product (IP) or further study observation. Note that the subject may need to undergo additional tests or tapering of treatment to withdraw safely, as applicable.
- Development of a serious or intolerable AE that necessitates discontinuation at the discretion of the Investigator (the AE section of the CRF/eCRF must be completed; AE includes serious adverse event (SAE) and death.
- 3. At the discretion of the Investigator, when he/she believes continued participation is not in the best interest of the subject.
- 4. At the discretion of the Investigator, when the subject does not adhere to the study procedures.
- 5. A protocol deviation that, in the opinion of the Sponsor and Investigator, warrants discontinuation from the study.

#### Lifestyle and/or Dietary Restrictions:

As defined in the inclusion and exclusion criteria, subjects are expected to follow lifestyle and dietary requirements.

| Investigational product, dose and mode of administration: |
|---|
| Name of Investigational Product 1: Fixed dose combination of olopatadine hydrochloride mug and |
| mometasone furoate µg NS |
| Manufacturing License Name: GSP 301 NS |
| Dosage Form: Spray, metered (Nasal Spray) |
| Dose: in each nostril |
| Dosage Frequency: |
| Mode of Administration: Intranasal |
| Placebo therapy, dosage and mode of administration: |
| Name: GSP 301 Placebo NS |
| Manufacturing License Name: GSP 301 Placebo NS |
| Dosage Form: Spray, metered (Nasal Spray) |
| Dosage: in each nostril |
| Dosage Frequency: |
| Mode of Administration: Intranasal |
| Duration of treatment: |
| Fourteen (14) days. |

#### Criteria for evaluation (see protocol section 13):

Study Endpoint(s)

#### Primary Endpoint

• Change from baseline in average AM and PM subject-reported 12-hour reflective Total Nasal Symptom Score (rTNSS) over the 14-day treatment period.

#### Secondary Endpoints:

In order of clinical importance (high to low), the secondary endpoints are as follows:

- Change from baseline in average AM and PM subject-reported 12-hour instantaneous Total Nasal Symptom Score (iTNSS) over the 14-day treatment period.
- Change from baseline in the overall Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) score on Day 15 (Visit 4) between treatment groups.
- Change from baseline in average AM and PM subject-reported 12-hour reflective Total Ocular Symptom Score (rTOSS) over the 14-day treatment period.

#### Other Efficacy Endpoints:

#### Nasal symptoms:

- Change from baseline in AM subject-reported rTNSS over the 14-day treatment period.
- Change from baseline in AM subject-reported iTNSS over the 14-day treatment period.
- Change from baseline in PM subject-reported rTNSS over the 14-day treatment period.
- Change from baseline in PM subject-reported iTNSS over the 14-day treatment period.
- Change from baseline in subject-reported reflective individual nasal symptoms over the 14-day treatment period (AM, PM, and average of AM and PM).
- Change from baseline in subject-reported instantaneous individual nasal symptoms over the 14-day treatment period (AM, PM, and average of AM and PM).
- Change from baseline in average AM and PM subject-reported rTNSS and iTNSS for each day.
- Change from baseline in AM subject-reported rTNSS and iTNSS for each day.
- Change from baseline in PM subject-reported rTNSS and iTNSS for each day.

#### Ocular symptoms:

- Change from baseline in average AM and PM subject-reported instantaneous Total Ocular Symptom Score (iTOSS) over the 14-day treatment period.
- Change from baseline in AM subject-reported rTOSS over the 14-day treatment period.
- Change from baseline in AM subject-reported iTOSS over the 14-day treatment period.
- Change from baseline in PM subject-reported rTOSS over the 14-day treatment period.
- Change from baseline in PM subject-reported iTOSS over the 14-day treatment period.
- Change from baseline in subject-reported reflective individual ocular symptoms over the 14-day treatment period (AM, PM, and average AM and PM).
- Change from baseline in subject-reported instantaneous individual ocular symptoms over the 14-day treatment period (AM, PM, and average AM and PM).
- Change from baseline in average of the AM and PM subject-reported rTOSS and iTOSS for each day.

- Change from baseline in AM subject-reported rTOSS and iTOSS for each day.
- Change from baseline in PM subject-reported rTOSS and iTOSS for each day.

Non-nasal symptoms will be assessed in a similar manner to the ocular symptoms above.

Physician assessed Nasal Symptom Score (PNSS):

Change from baseline in PNSS and physician assessed individual nasal symptoms at Day 15 (Visit 4).

Pediatric Rhinoconjuntivitis Quality of Life Questionnaire (PRQLQ):

• Change from baseline in individual domains of the PRQLQ at Day 15

#### Safety Endpoints

- AEs and SAEs.
- Vital signs.
- Physical examinations.
- Focused ears, nose, and throat (ENT)/Eye examinations.

#### Statistical methods:

Analysis Sets:

The Full Analysis Set (FAS) will consist of all subjects who have been randomized and received at least 1 dose of investigational product (IP) and have at least 1 post-baseline primary efficacy assessment. This will be the primary analysis set for efficacy analyses.

The Per Protocol Set (PPS) will consist of the subset of the FAS who do not meet criteria for PPS exclusion.

The Safety Analysis Set (SAS) will consist of all subjects who took at least 1 dose of study medication following randomization and will be used for all safety analyses.

Efficacy Analyses

The primary endpoint, change from baseline in average AM and PM subject-reported 12-hour rTNSS over a 14-day treatment period, will be evaluated using a mixed-effect repeated measures analysis of covariance (ANCOVA) model. The model will adjust for study treatment, site, baseline 12-hour rTNSS (linear, continuous covariate - defined as the average of the last 8 consecutive AM and PM assessments during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization) and study day as the within-subject effect, and site-by-treatment and baseline-by-treatment interactions. An unstructured variance-covariance matrix will be assumed as a start. Least square means of the treatment differences and associated 95% confidence intervals (CIs) and p-values will be presented. The primary analysis will be based on the FAS and a supportive analysis will be based on the PPS.

Analyses of the secondary and other endpoints will be performed using a similar method as described for the primary endpoint. Efficacy within pre-specified subgroups of clinical interest (eg, age, sex, race, and ethnicity) will be examined.

Primary and secondary efficacy endpoints will be analyzed using hierarchical testing in a fixed order. Treatment comparisons will begin with the primary endpoint versus placebo. If the resulting two-sided p-value is less than 0.05, then the next comparison of the secondary endpoint will be made, in the order of clinical importance. This process continues until either all comparisons of interest are made, or until the point at which the resulting two-sided p-value for a comparison of interest is greater than 0.05.

Safety Analyses

Descriptive statistics will be used to summarize AEs, vital signs, physical examination, focused ENT data and a comparison of the incidence rate of AEs between study drug groups will be presented.

Glenmark Specialty S.A.
Statistical Analysis Plan
Study Number - GSP 301-305

December 06, 2018

# TABLE OF CONTENTS

| 1. | LIST OF ABBREVIATIONS | 17 |
|---|---|---|
| 2. | INTRODUCTION | 20 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 21 |
| 3.1. | Study Objectives | 21 |
| 3.1.1 | Primary Objective | 21 |
| 3.1.2. | Secondary Objective | 21 |
| 3.2. | Study Endpoints | 21 |
| 3.2.1. | Primary Endpoint | 21 |
| 3.2.2. | Secondary Endpoints | 21 |
| 3.2.3 | Other Efficacy Endpoints | 21 |
| 3.2.4 | Safety Endpoints | 23 |
| 3.2.5 | Appropriateness of Measurements | 23 |
| 4. | STUDY DESIGN | 24 |
| 4.1. | Summary of Study Design | 24 |
| 4.2. | Definition of Study Drugs | 25 |
| 4.3. | Sample Size Considerations | 25 |
| 4.3.1. | Sample Size Justifications | 25 |
| 4.4. | Randomization | 26 |
| 4.5. | Clinical Assessments | 26 |
| 4.5.1. | Subject-Reported Nasal and Non-Nasal Symptoms | 26 |
| 4.5.2. | Pediatric Rhinoconjunctivitis Quality-Of-Life Questionnaire (PRQLQ) | 27 |
| 4.5.3. | Physician Assessed Nasal Symptom Score (PNSS) | 28 |
| 5. | PLANNED ANALYSES | 29 |
| 5.1. | Interim Analyses | 29 |
| 5.2. | Final Analyses | 29 |
| 6. | GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING | 30 |
| 6.1. | General Summary Table and Individual Subject Data Listing Considerations | 30 |
| 6.2. | General Post Text Summary Table and Individual Subject Data Listing Format Considerations | 30 |
| 6.3. | Data Management | 30 |

| ottidy IN | umber - (13) 301-305 | ciliber ob, 2018 |
|---|---|---|
| 6.4. | Data Presentation Conventions | 31 |
| 6.5. | Analysis Populations | 32 |
| 6.5.1. | Run-In Set | 32 |
| 6.5.2. | Full Analysis Set (FAS) | 32 |
| 6.5.3. | Per Protocol Set (PPS) | 32 |
| 6.5.4. | Safety Analysis Set (SAS) | 32 |
| 6.6. | Baseline Definition | 33 |
| 6.7. | Derived and Transformed Data | 33 |
| 6.7.1. | Baseline Age | 33 |
| 6.7.2. | Study Day | 34 |
| 6.7.3. | Change from Baseline | 34 |
| 6.7.4. | Visit Windows | 34 |
| 6.7.5. | Unscheduled Visits | 35 |
| 6.8. | Handling of Missing Data | 35 |
| 6.8.1. | Missing Efficacy Endpoints | 35 |
| 6.8.2. | Missing Start and Stop Dates for Prior and Concomitant Medication | 35 |
| 6.8.3. | Missing Start and Stop Dates for Adverse Events | 35 |
| 7. | STUDY POPULATION | 36 |
| 7.1. | Subjects Disposition | 37 |
| 7.2. | Protocol Deviations | 37 |
| 7.3. | Demographic and Baseline Characteristics | 37 |
| 7.4. | Listing of Subject Inclusion and Exclusion Criteria | 37 |
| 7.5. | Medical History and Medical Conditions Present at Entry | 37 |
| 7.6. | Prior Medication History and Medications Present at Entry | 38 |
| 7.7. | Baseline Physical Examination | 38 |
| 7.8. | Baseline Vital Signs | 38 |
| 7.9. | Baseline Focused ENT/Eye examination | 38 |
| 7.10. | Baseline Efficacy Evaluations | 38 |
| 8. | EFFICACY | 40 |
| 8.1. | General Considerations | 40 |
| 8.2. | Statement of the Null and Alternate Hypotheses | 40 |
| 8.3. | Subgroup Analyses | 41 |

| Statistical A | Specialty S.A. Analysis Plan ber - GSP 301-305 December 06, 2018 | |
|---|---|---|
| 8.4. | Multiple Comparisons and Multiplicity4 | 1 |
| 8.5. | Analysis of the Primary Efficacy Endpoint | |
| 8.5.1. | Primary Efficacy Analysis4 | |
| 8.6. | Analysis of the Secondary Efficacy Endpoints4 | |
| 8.6.1. | Analysis of Change from Baseline in iTNSS and rTOSS4 | |
| 8.6.2. | Analysis of Change from Baseline in the Overall PRQLQ on Day 154 | |
| 8.7. | Efficacy Analyses of Other Endpoints of Interest4 | 5 |
| 8.8. | Summary of Reasons for Efficacy Non-Evaluability/Exclusion from Efficacy Analyses | |
| 9. | SAFETY AND TOLERABILITY4 | 7 |
| 9.1. | Overall Summary of Tolerability4 | 7 |
| 9.2. | Adverse Event Preferred Term and Body/Organ System Summary Tables4 | 8 |
| 9.2.1. | Summaries of Adverse Event Incidence Rates for All Subjects4 | 8 |
| 9.2.2. | Missing and Partial AE Dates4 | 8 |
| 9.2.3. | Summaries of Adverse Incidence Rates for Serious Adverse Events (SAE), adverse events leading to discontinuation, and treatment-related emergent adverse events | 0 |
| 9.3. | Total Duration of Therapy, Average Daily Dose, Maximum Daily Dose, Final Daily Dose of Study Medication, treatment Compliance and diary compliance | 0 |
| 9.4. | Concomitant and Other Medications5 | 1 |
| 9.4.1. | Missing and Partial Concomitant and Other Medication Start and Stop Dates5 | 1 |
| 9.5. | Pregnancy Test5 | 1 |
| 9.6. | Vital Signs5 | 1 |
| 9.7. | Physical Examination5 | 2 |
| 9.8. | Focused ENT/Eye examination | 2 |
| 9.9. | Study Termination Status5 | 3 |
| 10. | CHANGES IN ANALYSES FROM THE PROTOCOL5 | 4 |

11.

REFERENCES ......55

# LIST OF TABLES

| Table 1: | List of Abbreviations | 17 |
|----------|-------------------------------------------------------|----|
| Table 2: | Visit Windows (Days) | 34 |
| Table 3: | Overview of Planned Study Population Analyses | 36 |
| Table 4: | Overview of Efficacy Analysis of the Primary Endpoint | 40 |
| Table 5: | Overview of Planned Secondary Efficacy | 43 |
| Table 6: | Overview of Planned Safety Analyses | 47 |
| Table 7: | Normal ranges of vital signs | 52 |

# 1. LIST OF ABBREVIATIONS

**Table 1:** List of Abbreviations

| Abbreviation | Definition or Explanation |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse event |
| AM | Morning (ante meridian, before noon) |
| ANCOVA | Analysis of covariance |
| AR | Allergic rhinitis |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CRF | Case report form |
| CRO | Contract research organization |
| CSR | Clinical study report |
| DV | Discontinuation visit |
| eCRF | Electronic case report form |
| ENT | Ears, nose, and throat |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration (of the United States) |
| FDC | Fixed dose combination |
| GSP 301 NS | NS Fixed dose combination of olopatadine hydrochloride and mometasone furoate nasal spray |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| iTNSS | Instantaneous Total Nasal Symptom Score |

| Abbreviation | Definition or Explanation |
|---|---|
| iTNNSS | Instantaneous Total Non-Nasal Symptom Score |
| iTOSS | Instantaneous Total Ocular Symptom Score |
| IVRS | Interactive Voice Response System |
| IWRS | Interactive Web Response System |
| J2R | Jump to Reference |
| LSM | Least squares mean |
| μg | microgram |
| MAR | Missing at random |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed-effect Model Repeated Measures |
| MNAR | Missing not at random |
| NS | Nasal spray |
| OTC | Over-the-counter |
| PM | Evening |
| PNSS | Physician Assessed Nasal Symptom Score |
| PPS | Per protocol set |
| PRQLQ | Pediatric Rhinoconjunctivitis Quality of Life Questionnaire |
| PT | Preferred term |
| rTNSS | Reflective Total Nasal Symptom Score |
| rTNNSS | Reflective Total Non-Nasal Symptom Score |
| rTOSS | Reflective Total Ocular Symptom Score |
| RV | Randomization visit |
| SAE | Serious adverse events |
| SAP | Statistical analysis plan |
| SAR | Seasonal allergic rhinitis |
| SAS | Safety analysis set |
| SD | Standard deviation |

| SDTM | Study Data Tabulation Model |
|-------|----------------------------------|
| SOC | System organ class |
| SPT | Skin Prick Test |
| SV | Screening visit |
| TEAE | Treatment-emergent adverse event |
| TNSS | Total Nasal Symptom Score |
| TNNSS | Total Non-Nasal Symptom Score |
| TOSS | Total Ocular Symptom Score |
| TV | Treatment visit |
| US | United States |
| VS | Versus |

#### 2. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide details of the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures to be included in the Clinical Study Report (CSR) for Protocol GSP 301-305.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

| Clinical Study Protocol<br>(Study No. GSP 301-305) | 08-JAN-2018 | Version 1.0 |
|---|---|---|
| Clinical Study Protocol Amendment 1 (Study No. GSP 301-305) | 05-APR-2018 | Version 2.0 |
| GSP 301-305 Subject Case Report Forms | 12-MAR-2018 | Version 1.0 |

This SAP was developed in accordance with ICH E9 guideline. The document may evolve over time, for example, to reflect the requirements of protocol amendments or regulatory requests. However, the final SAP must be finalized, approved by the Sponsor, and placed on file before database is locked. Deviations from the final approved plan will be noted in the clinical study report. Further information can be found in the clinical study protocol.

The protocol states that the primary endpoint will be evaluated using a repeated measures analysis of covariance (ANCOVA) model. The terminology mixed-effect model repeated measures (MMRM) model will be applied throughout the SAP instead of repeated measures ANCOVA for precision.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

## 3.1.1. Primary Objective

To compare the efficacy of GSP 301 NS (administered as over 14 days of study drug in pediatric subjects (aged ≥6 to <12 years) with SAR.

#### 3.1.2. Secondary Objective

To assess the safety and tolerability over 14 days of study drug in pediatric subjects (aged  $\geq$ 6 to <12 years) with SAR.

# 3.2. Study Endpoints

#### 3.2.1. Primary Endpoint

• Change from baseline in average AM and PM subject-reported 12-hour reflective Total Nasal Symptom Score (rTNSS) over the 14-day treatment period.

#### 3.2.2. Secondary Endpoints

In order of clinical importance (high to low), the secondary endpoints are as follows:

- Change from baseline in average AM and PM subject-reported 12-hour instantaneous Total Nasal Symptom Score (iTNSS) over the 14-day treatment period.
- Change from baseline in the overall Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) score on Day 15 (Visit 4) between treatment groups.
- Change from baseline in average AM and PM subject-reported 12-hour reflective Total Ocular Symptom Score (rTOSS) over the 14-day treatment period.

#### 3.2.3. Other Efficacy Endpoints

Nasal symptoms:

- Change from baseline in AM subject-reported rTNSS over the 14-day treatment period.
- Change from baseline in AM subject-reported iTNSS over the 14-day treatment period.
- Change from baseline in PM subject-reported rTNSS over the 14-day treatment period.
- Change from baseline in PM subject-reported iTNSS over the 14-day treatment period.
- Change from baseline in subject-reported reflective individual nasal symptoms over the 14-day treatment period (AM, PM, and average of AM and PM).

- Change from baseline in subject-reported instantaneous individual nasal symptoms over the 14-day treatment period (AM, PM, and average of AM and PM).
- Change from baseline in average AM and PM subject-reported rTNSS and iTNSS for each day.
- Change from baseline in AM subject-reported rTNSS and iTNSS for each day.
- Change from baseline in PM subject-reported rTNSS and iTNSS for each day.

#### Ocular symptoms:

- Change from baseline in average AM and PM subject-reported instantaneous Total Ocular Symptom Score (iTOSS) over the 14-day treatment period.
- Change from baseline in AM subject-reported rTOSS over the 14-day treatment period.
- Change from baseline in AM subject-reported iTOSS over the 14-day treatment period.
- Change from baseline in PM subject-reported rTOSS over the 14-day treatment period.
- Change from baseline in PM subject-reported iTOSS over the 14-day treatment period.
- Change from baseline in average of the AM and PM subject-reported rTOSS and iTOSS for each day.
- Change from baseline in AM subject-reported rTOSS and iTOSS for each day.
- Change from baseline in PM subject-reported rTOSS and iTOSS for each day.

Please note that the individual ocular symptoms are part of the Non-nasal Symptoms. As such, summary tables will be produced and will be found for each of these individual symptoms only under the Non-nasal Symptoms title (will not repeat under TOSS).

#### Non-nasal symptoms:

- Change from baseline in average AM and PM subject-reported instantaneous Total Non-Nasal Symptom Score (iTNNSS) over the 14-day treatment period.
- Change from baseline in average AM and PM subject-reported reflective Total Non-Nasal Symptom Score (rTNNSS) over the 14-day treatment period.
- Change from baseline in AM subject-reported rTNNSS over the 14-day treatment period.
- Change from baseline in AM subject-reported iTNNSS over the 14-day treatment period.

- Change from baseline in PM subject-reported rTNNSS over the 14-day treatment period.
- Change from baseline in PM subject-reported iTNNSS over the 14-day treatment period.
- Change from baseline in subject-reported reflective individual non-nasal symptoms over the 14-day treatment period (AM, PM, and average AM and PM).
- Change from baseline in subject-reported instantaneous individual non-nasal symptoms over the 14-day treatment period (AM, PM, and average AM and PM).
- Change from baseline in average of the AM and PM subject-reported rTNNSS and iTNNSS for each day.
- Change from baseline in AM subject-reported rTNNSS and iTNNSS for each day.
- Change from baseline in PM subject-reported rTNNSS and iTNNSS for each day.

Physician assessed Nasal Symptom Score (PNSS):

• Change from baseline in PNSS and physician assessed individual nasal symptoms at Day 15 (Visit 4).

Pediatric Rhinoconjuntivitis Quality of Life Questionnaire (PRQLQ):

• Change from baseline in individual domains of the PRQLQ at Day 15.

## 3.2.4. Safety Endpoints

- AEs and serious adverse events (SAEs).
- Vital signs.
- Physical examinations.
- Focused ears, nose, and throat (ENT)/Eye examinations.

#### 3.2.5. Appropriateness of Measurements

The change in the rTNSS as a primary endpoint and the treatment duration of 14 days is per the FDA guidance, "Allergic Rhinitis: Developing Drug Products for Treatment – Guidance for Industry (Draft Guidance)", as well as similar previously published studies.

The safety assessments to be performed in this study, including assessment of AEs, vital signs, physical examination are standard evaluations to ensure subject safety.

#### 4. STUDY DESIGN

# 4.1. Summary of Study Design

This is a randomized, double-blind, parallel-group, placebo-controlled comparative study to evaluate the efficacy and safety of GSP 301 NS administered as compared with GSP 301 placebo NS at the same dose and in the same vehicle in subjects with seasonal allergic rhinitis (SAR). Subjects will be enrolled during the spring or fall allergy seasons and will be randomized to treatment in a 1:1 ratio to the following two treatment groups, at multiple study sites:

- GSP 301 NS μg olopatadine hydrochloride μg mometasone furoate administered as
- GSP 301 placebo NS

The placebo used in the study are formulated in the same vehicle as GSP 301 NS and all the NS bottles are identical in appearance. Thus, other than the active component of each treatment, there are no other differences in the formulation or the bottle of each treatment.

Pollen counts will be obtained each weekday, and when possible, each weekend day at each investigational site, either by study staff or by a community counting station located within approximately 30 miles of the study site. Three (3) consecutive days of moderate pollen counts will be accepted as the start to that pollen's given allergy season. Pollen counts will be entered as part of the data entry in the CRFs/eCRFs or other methods as provided by the Sponsor or designee.

This study consists of 4 visits to the study site (Figure 1). After the initial Screening Visit (Visit 1), subjects who meet all study selection criteria will undergo a single blind, placebo, run-in period for 7 to 10 days. Following the completion of run-in period, eligible subjects meeting the randomization criteria will be enrolled and randomized to 1 of the 2 treatment groups. Randomized subjects will undergo a 2-week (14-day) treatment period to assess the efficacy and safety of the assigned treatment.

No scheduled post-treatment follow-up visit is planned for this study. However, if the subject is withdrawn because of an AE, the AE will be followed until the medical condition returns to baseline or is considered stable or chronic. If needed, additional unscheduled visits/telephone visits may be conducted at any time during the study to ensure subject safety or to perform other study-related procedures at the discretion of the Investigator or the Sponsor.

Figure 1: Study Design Schematic



# 4.2. Definition of Study Drugs

Name of Investigational Product: FDC of olopatadine hydrochloride µg and mometasone furoate µg NS (GSP 301 NS)
License Name: GSP 301 NS
Dosage Form: NS
Dosage: in each nostril
Dosage Frequency: for 14 days
Mode of Administration: Intranasal

Reference Product: GSP 301 placebo NS License Name: GSP 301 placebo NS

Dosage Form: NS

Dosage: in each nostril

Dosage Frequency: for 14 days

Mode of Administration: Intranasal

GSP 301 placebo NS is the reference product with pH 3.7 and will be referred to throughout this document as "placebo NS".

The study medication will be dispensed at the study site after adequate training using a placebo NS bottle.

# 4.3. Sample Size Considerations

#### 4.3.1. Sample Size Justifications

A total sample size of 450 randomized subjects (225 subjects per treatment group) has been selected for this study.

The primary goal of the analysis of the primary endpoint will be to assess the superiority of GSP 301 NS versus (vs) GSP 301 placebo NS.

A sample size of 382 evaluable subjects, allocated 1:1, will provide 90% power to detect a between-group mean difference (GSP 301 NS vs placebo NS) of 1.0 in the absolute change from baseline in average AM and PM subject-reported 12-hour rTNSS over a 14-day treatment period (assuming a two-sided alpha of 5%). A standard deviation of 3.0 in the change from baseline in 12-hour rTNSS over a 14-day treatment period has been assumed. Assuming a drop-out rate of 15%, a total of approximately 450 subjects are planned to be randomized (225 subjects in each treatment group). Depending on the actual drop-out rate, the sponsor may decide to randomize high or lower number of subjects in order to meet the required sample size of 382 evaluable subjects.

## 4.4. Randomization

Subjects will be assigned to 1 of the 2 treatment groups in a 1:1 ratio based on a computer-generated randomization scheme that will be reviewed and approved by a statistician. The randomization will be performed centrally using IVRS/IWRS. The randomization scheme and treatment allocation for each subject will be included in the final clinical study report (CSR) for this study.

This study is designed as a double-blind study. The blinding will be maintained by packing the active products and placebo in identical bottles and outer cartons. Double-blind kits containing the IP will be supplied to the sites and will be dispensed to subjects using IVRS/IWRS.

#### 4.5. Clinical Assessments

## 4.5.1. Subject-Reported Nasal and Non-Nasal Symptoms

#### Nasal Symptoms

The primary efficacy measure in this study is the subject-reported TNSS. The TNSS is defined as the sum of the subject-reported symptom scores for four nasal symptoms: rhinorrhea (runny nose), nasal congestion, nasal itching, and sneezing. The subject will assess and report his/her nasal symptoms twice (in morning [AM assessment] and evening [PM assessment]) on each day of the placebo run-in and double-blind treatment periods prior to administering the study treatment. If a nasal symptom score is missing, then the TNSS will be set to missing.

The subject will be asked to assess both reflective (i.e. an evaluation of symptom severity over the past 12 hours prior to the recording of the score) and instantaneous nasal symptoms (i.e evaluation of the symptom severity just before taking study medication [within 10 minutes]).

Each of the following symptoms will be assessed.

| Nasal Symptoms | |
|-----------------------------------|-------------|
| 1. Nasal Congestion 2. Rhinorrhea | |
| 3. Nasal Itching | 4. Sneezing |

Each of the above symptoms will be rated on a 4-point scale as follows:

| | Grade | Description |
|---|---|---|
| 0 | Absent | No Sign/Symptoms evident |
| 1 | Mild | Sign/Symptoms clearly present but minimal awareness; easily tolerated |
| 2 | Moderate | Definite awareness of sign/symptoms which is bothersome but tolerable |
| | | Sign/symptoms is hard to tolerate; causes interference with activities of |
| | | daily living and or sleeping |

#### Non-Nasal Symptoms

The efficacy measures in this study will also include the subject-reported Total Non-nasal Symptom Score. The Total Non-nasal Symptom Score is defined as the sum of the subject reported non-nasal symptom scores for four non-nasal symptoms: itching/burning eyes, tearing/watering eyes, redness of eyes, and itching of ears or palate. The subject will assess and report his/her non-nasal symptoms twice (in morning [AM assessment] and evening [PM assessment]) on each day of the placebo run-in and treatment periods prior to administering the study treatment. If a non-nasal symptom score is missing, then the total non-nasal symptom score will be set to missing.

The subject will be asked to assess both reflective (i.e., an evaluation of symptom severity over the past 12 hours prior to the recording of the score) and instantaneous (evaluation of the symptom severity just before taking study medication [within 10 minutes]).

Each of the following symptoms will be assessed.

| Non-Nasal Symptoms | |
|---|---|
| 1. Itching/ Burning Eyes 2. Tearing/ Watering Eyes | |
| 3. Redness of Eyes | 4. Itching of Ears or Palate |

Each of the above symptoms will be rated on a 4-point scale as follows:

| | Grade | Description |
|---|---|---|
| 0 | Absent | No Sign/Symptoms evident |
| 1 | Mild | Sign/Symptoms clearly present but minimal awareness; easily tolerated |
| 2 | Moderate | Definite awareness of sign/symptoms which is bothersome but |
| | | tolerable |
| 3 | Severe | Sign/symptoms is hard to tolerate; causes interference with activities |
| | | daily living and or sleeping |

The Total Ocular Symptom Score (TOSS) will be calculated using the 3 eye-related non-nasal symptoms - itching/burning eyes, tearing/watering eyes, and redness of eyes. If an eye-related non-nasal symptom score is missing, then the TOSS will be set to missing.

# 4.5.2. Pediatric Rhinoconjunctivitis Quality-Of-Life Questionnaire (PRQLQ)

The PRQLQ used in this study is a validated, disease-specific, quality-of-life questionnaire developed to measure the physical, emotional, and social impairments that are experienced by children (age  $\geq 6$  to < 12 years) with rhinoconjunctivitis. The PRQLQ has 23 questions in 5

domains (nose symptoms, eye symptoms, practical problems, activity limitation and other symptoms). Subjects will be asked to recall their experiences during the previous week and to give their responses on a 7-point scale.

PRQLQ scores will be summarized by domains. A domain average score is calculated as the sum of the scores in that domain divided by the number of items in that domain; all items in the domain must be valid in order to calculate the corresponding average score. A domain average score will be set to missing if there is a missing item score in that domain.

The overall average PRQLQ score is calculated as the sum of the scores in all domains divided by the total number of items in the five domains; all items in the 5 domains must be valid in order to calculate the corresponding overall average score. If a domain score is missing, then the overall average PRQLQ score will be set to missing.

## 4.5.3. Physician Assessed Nasal Symptom Score (PNSS)

The Physician-Assessed Total Nasal Symptom Score (PNSS) will be derived from the intensity of the following nasal symptoms associated with AR - rhinorrhea (runny nose), nasal congestion, nasal itching, and sneezing. Physicians will assess severity of the above symptoms for subject-reported nasal symptoms. The severity grading is a 4-point scale similar to other assessments (0-absent, 1-mild, 2-moderate, 3-severe). The PNSS will be based on questioning of the subjects (overall feeling since last visit) and on the ENT examination and other observations by the physician. If a nasal symptom is missing, then the PNSS will be set to missing.

## 5. PLANNED ANALYSES

# 5.1. Interim Analyses

There is no interim analysis planned in this study.

# 5.2. Final Analyses

All planned analyses will be carried out once the clinical database lock (DBL) has taken place. Once this has been achieved, unblinding will occur and the analyses will be performed.

# 6. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING

# 6.1. General Summary Table and Individual Subject Data Listing Considerations

In general, listings will be sorted and presented by treatment and subject number. Subject number when broken down consists of the Site Number and Subject Number. Randomization number will be included in listing of demographic data. Study visits will be labeled as Screening, Baseline, Day 8 and Day 15.

The following treatment labels will be used for all tables, figures and listings in the order below:

| Placebo NS |
|------------|
| GSP 301 NS |

# 6.2. General Post Text Summary Table and Individual Subject Data Listing Format Considerations

Tables, Listings and Figures are numbered following the ICH structure. No gaps are to be in the table, figure and listing output numbering (e.g. 14.1.1, 14.1.2, 14.1.3). Table headers, variables names and footnotes will be modified as needed following data analyses. Additional Tables, Listings and Figures will be generated, as needed, following the data analysis (post-hoc).

# 6.3. Data Management

Data from the study will be managed by the Sponsor's Clinical Research Operations group or designee. A copy of the study results will be made available to the Clinical Investigator for review.

All data will be directly recorded on the CRFs/eCRFs. The Investigator will allow representatives of the Sponsor, regulatory agencies, and their designees to inspect all study documents (including, but not limited to, consent forms, IP accountability forms, IRB/IEC approvals) and pertinent hospital or clinic records for confirmation of data throughout and after completion of the study. Monitoring visits will be conducted as needed during the course of the study. A complete review of source documentation of key efficacy and safety data will be conducted at each monitoring visit for verification that all information recorded in the CRF/eCRF accurately reflects the data recorded in the subject's source documents.

All data verification, using hospital or clinic records, will be performed respecting subject confidentiality and will be carried out in accordance with SOPs.

All subject data generated during the study will be recorded and transcribed into a database. The Principal Investigator must approve the CRF/eCRF to confirm eligibility. The final authorization of the CRF/eCRF data is the Investigator Signature Form. This form must be approved by the Principal Investigator to signify that he/she has reviewed the CRF/eCRF, including all laboratory and safety assessments, and that all of the data therein is complete and accurate.

The data will be reviewed to ensure that the forms were completed properly.

Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4, unless otherwise noted.

#### 6.4. Data Presentation Conventions

Few important highlights as well as other important specifications are included here:

• The following conventions are applied to all data presentations and summaries:

## o Descriptive statistics

Minimum, Maximum: the same number of decimal places as the raw data Arithmetic mean, Standard Deviation (SD), Median: 1 more decimal place than the raw data.

Descriptive statistics will be presented aligned by decimal point.

#### o Categorical Variables

The number and percentage of the responses are presented in the form xxx (xx.x)

Percentages: 1 decimal place

No display of percentage in case that number of subject is zero unless otherwise stated

#### o P-values

3 decimal places

If the p-value is less than 0.001 then it will be presented as <0.001. If the rounded result is a value of 1.000, it will be displayed as >0.999

## o Confidence Interval (CI) limits

The same decimal places as the estimate (in the case of mean, 1 more decimal place than the raw data, and in the case of percentage, 1 decimal place)

- A table, figure, listing is to be generated for any required item where no data is available or reported. This will ensure to the health authorities that the tables, figures, listings and narratives are accounted for.
  - Generate a table or listing which states "No Data Available" or "No Data Reported"
  - Print a one-line message indicating there was no report data available: "NO DATA AVAILABLE FOR THIS REPORT"

# 6.5. Analysis Populations

#### 6.5.1. Run-In Set

The Run-In Analysis Set will consist of subjects enrolled in placebo run-in period (between the subjects signing informed consent and administration of the first dose of the randomized study medication) and will be used for presenting run-in period AEs, concomitant medication and protocol deviations.

## 6.5.2. Full Analysis Set (FAS)

The FAS will consist of all subjects who are randomized and received at least one dose of investigational product and have at least one post-baseline primary efficacy assessment. If a subject is randomized in the study more than one time, it will be decided at the Blind Data Review Meeting (BDRM) on a case by case basis if the subject should be included in FAS. Full analysis set will be the primary analysis set for efficacy analyses.

#### 6.5.3. Per Protocol Set (PPS)

The PPS will consist of the subset of the FAS who do not meet criteria for PPS exclusion. These criteria are to capture relevant non-adherence to the protocol (defined as a 'major deviation', especially those that affect interpretation of the primary endpoint). The PPS will be a secondary analysis set for the primary and secondary efficacy endpoints, except for PRQLQ which will be performed only on FAS. The PPS will be used to assess the robustness of the results from the statistical tests based on the FAS.

Major deviations will lead to the exclusion of a subject from the PPS. Major protocol deviations will be identified during the Blinded Data Review Meeting (BDRM) before database lock. Major protocol deviations *may* include:

- Subjects who had their blinded randomization code broken.
- Subjects with overall treatment compliance <75% or >125%.
- Subjects who used prohibited medications (prior and/or concomitant) that may have significant influence on efficacy.
- Subjects who did not satisfy the inclusion/exclusion that may have significant influence on efficacy.
- Subjects not treated with the treatment assigned at randomization, but wrongly treated in another treatment group.

#### 6.5.4. Safety Analysis Set (SAS)

The Safety Analysis Set (SAS) will consist of all subjects who are randomized and receive at least one dose of study medication following randomization and will be used for all safety analyses.

#### 6.6. Baseline Definition

Unless otherwise specified, the following general principles apply for determining the baseline for daily diary variables and for variables collected during scheduled visits:

## Primary endpoint parameter rTNSS

The baseline will be defined as the average of the last 8 consecutive AM and PM assessments during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization. At least 6 out of 8 reading scores should be available in order to calculate baseline score.

## Secondary and other 12-hour average AM and PM endpoint parameters

The same method will be used to determine the baseline for secondary and other 12-hour average AM and PM efficacy endpoint parameters:

- average AM and PM rTNSS, iTNSS, and corresponding AM and PM individual symptoms
- average AM and PM rTOSS; average AM and PM iTOSS
- average AM and PM rTNNSS, average AM and PM iTNNSS and corresponding individual symptoms

## Other endpoints for AM or PM nasal/non-nasal symptoms

The baseline score will be defined as the average of the last 4 consecutive AM or PM assessments (respectively for either AM or PM corresponding endpoint) during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization. At least 3 out of 4 reading scores should be available in order to calculate baseline score.

#### Safety endpoints

Unless otherwise specified, 'baseline' for safety analysis will be defined as the last available assessment prior to the first dose of study drug following randomization.

#### PROLO and PNSS

Baseline is defined as the score at the Randomization Visit (Day 1; Visit 2).

### 6.7. Derived and Transformed Data

#### 6.7.1. Baseline Age

Age is the subject's age in years calculated based on the informed consent date and subject's date of birth.

If the month and day of informed consent is on or after the month and day of birth:

Age = year of informed consent - year of birth

If the month and day of informed consent is before the month and day of birth:

Age = year of informed consent – year of birth – 1

## 6.7.2. Study Day

If the date of interest occurs on or after the randomization date:

Study day = date of interest - randomization date + 1

If the date of interest occurs before the randomization date:

Study day = date of interest - randomization date

There is no study day 0.

# 6.7.3. Change from Baseline

Change from baseline in average AM and PM 12-hour rTNSS over a 14-day treatment period

- For mixed-effect model repeated measures (MMRM) model, this will be derived by calculating a mean score for each subject, based on the post-dose PM of the dosing day and AM assessment of next day for each day (ie Day 1 measurement = Average of the PM assessment on Day 1 and AM assessment of Day 2 and so on).
- For Analysis of Covariance (ANCOVA) model, the overall mean change from baseline over the 14 day period includes assessment from Day 1 PM assessment through Day 15 in the morning.

The same derivation method will be applied to endpoint change from baseline in average AM and PM 12-hour for iTNSS, rTOSS, iTOSS, rTNNSS, iTNNSS, individual reflective/instantaneous nasal/non-nasal symptom scores.

For all other endpoints, change from baseline is calculated as the difference between the post-baseline result and the baseline result.

Percent change is calculated as (change from baseline / baseline result \* 100).

#### 6.7.4. Visit Windows

Subject participation may be 22 days up to 27 days with 7 to 10 days of a screening/run-in period and a 14-day treatment period, with allowable window periods for the study visits. The following visit windows are permitted: ±2 days for the Treatment Visit (Visit 3) and +2 days for the Final Visit/Discontinuation Visit (Visit 4). However, only data up to Day 15 AM is to be included in the efficacy analysis of subject-reported nasal and non-nasal symptoms.

Table 2: Visit Windows (Days)

| Visit | Relative Target Day | Visit Window |
|---------------------------------|---------------------|--------------|
| Visit 1 (Screening) | <i>-</i> 7 | -107 |
| Visit 2 (Randomization) | 1 | 1 |
| Visit 3 (Treatment) | 8 | 6-10 |
| Visit 4 (Final/Discontinuation) | 15 | 15 – 17 |

#### 6.7.5. Unscheduled Visits

An unscheduled visit (or telephone follow-up) may be performed at any time during the study at the subject's request or as deemed necessary by the Investigator. The date and reason for the unscheduled visit will be recorded on the CRF/eCRF as well as any other data obtained (eg, AEs, concomitant medications/treatments, and results from procedures or tests).

Data collected at unscheduled visits will be included in the listings, but not in the summary tables.

# 6.8. Handling of Missing Data

## 6.8.1. Missing Efficacy Endpoints

- Change from baseline in average AM and PM 12-hour rTNSS over a 14-day treatment period: For mixed-effect model repeated measures (MMRM) model if an AM or PM measurement is missing then the non-missing AM or PM measurement is used as the mean response for that day. If both the AM and PM measurement is missing then the mean response for that day will be missing.
  - The same methodology will be applied to endpoints of change from baseline in average AM and PM 12-hour iTNSS, rTOSS, iTOSS, rTNNSS, iTNNSS, individual reflective/ instantaneous nasal/non-nasal symptom scores.
- If either the baseline or the post-baseline result is missing, the change from baseline and percent change are also set to missing.

# 6.8.2. Missing Start and Stop Dates for Prior and Concomitant Medication

See section 9.4.

#### 6.8.3. Missing Start and Stop Dates for Adverse Events

See section 9.2.
#### 7. STUDY POPULATION

The study population analyses will be based on the safety analysis set, unless otherwise specified. Table 3 provides an overview of the planned study population analyses.

Table 3: Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject disposition | | | |
| Total screened | Y[1] | | |
| Treated with study medication during run-in period | Y[1] | | |
| Randomized | Y[2] | | |
| Study completion/withdrawal | Y[2] | | Y |
| Reason for early termination | Y[2] | | Y |
| Protocol Deviations | | | |
| Protocol deviations during randomized treatment period | Y[2] | | Y |
| Protocol deviations during run-in period | Y[2] | | Y |
| Protocol deviations during pre-run-in period | Y[1] | | Y |
| Major protocol deviations | Y[2] | | Y[4] |
| Subjects included in /excluded from analysis populations | | | |
| Summary of subjects in analysis population | Y[2] | | |
| Subjects excluded from each analysis populations | | | Y |
| Subjects who withdrew due to inclusion/exclusion | | | Y |
| criteria with criteria number and description | | | Y |
| Demographic and Baseline Characteristics | | | Ni<br>Ur |
| Demographic Characteristics | Y[3] | | Y |
| Skin Prick Test/Allergy Testing | | | Y |
| Medical History | | | Y |
| Exposure and Treatment and Diary Compliance | | | |
| Exposure during randomized treatment period | Y[2] | | Y |
| Treatment Compliance during randomized treatment period | Y[2] | | Y |
| Diary Compliance | | | Y |
| Concomitant Medications | | | |
| Prior Medications | | | Y |
| Concomitant Medications during randomized treatment | | | |
| period | | | Y |
| Concomitant Medications during run-in period | | | Y |
| Pollen Count and Rain Data | | | |
| Pollen and rain count listing by site | | | Y |
| NOTES: | | | |

#### NOTES:

- Y = Yes display generated
- [1]: Data from clinic or database
- [2]: Display will be based on the SAS

| Display Type | Data D | Data Displays Generate | |
|--------------|--------|------------------------|---------|
| | Table | Figure | Listing |

- [3]: Display will be based on the SAS population and repeated for the FAS and PPS populations
- [4]: Major protocol deviations will be included in the listings of all protocol deviations.

#### 7.1. Subjects Disposition

The subject accountability and disposition information will be summarized by study treatment group. The number of subjects screened, treated with study medication during the run-in period, randomized, treated with study medication following randomization, and the number of subjects in each analysis set will be tabulated. In addition, completion status and primary reason for withdrawal will be summarized by study treatment group.

#### 7.2. Protocol Deviations

Important protocol deviations (PDs) will be listed and summarized by study treatment group, separately for pre-run-in, run-in and randomized treatment periods. Major deviations will lead to patients being excluded from the per-protocol analysis set as defined in Section 6.5.3. Major protocol deviations will be listed and discussed in the CSR.

#### 7.3. Demographic and Baseline Characteristics

Subject demographic information will be collected at the Screening Visit (Visit 1). Demographic information includes age sex, race/ethnicity, will be summarized by treatment group separately for the SAS, FAS, and PPS analysis set. Other baseline characteristics including allergen test will be displayed in listing.

Continuous variables such as age will be summarized using descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum). Categorical variables such as sex and race will be summarized using frequencies and percentage.

All data will be listed by treatment and subject.

## 7.4. Listing of Subject Inclusion and Exclusion Criteria

All patients who failed any inclusion/exclusion criteria will be listed along with details of the failed criteria.

Failed inclusion/exclusion data will be listed by treatment and subject.

#### 7.5. Medical History and Medical Conditions Present at Entry

All relevant medical and surgical history and current medical conditions will be recorded at the Screening Visit (Visit 1).

Medical history data will be listed by treatment and subject.

#### 7.6. Prior Medication History and Medications Present at Entry

At Visit 1 subjects will be questioned about prior medication history and medications present at entry. Prior medications are defined as medications that started and ended before the first administration of the study medication.

All prior medications taken will be listed by treatment and subject.

#### 7.7. Baseline Physical Examination

Physical examinations (comprehensive) will be performed at the Screening Visit (Visit 1).

Descriptive statistics (frequency and percentage) will be used to summarize physical examination results by body system, treatment group and visit. In addition, the number of subjects with values of potential clinical significance determined by the investigator will be tabulated.

All physical examination data will be listed by treatment and subject.

#### 7.8. Baseline Vital Signs

The subject's baseline vital signs will be recorded (pulse rates, sitting systolic and diastolic blood pressure, height and weight) at Randomization Visit (Visit 2). Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be used to summarize vital sign results by treatment group and visit.

Values outside the respective normal range and values deemed as clinically significant by the Investigator will be listed.

The number of subjects with values of potential clinical significance determined by the investigator will be tabulated by treatment group and visit.

#### 7.9. Baseline Focused ENT/Eye examination

The subject's baseline focused ENT/Eye examinations will be performed at Randomization Visit (Visit 2). Descriptive statistics (frequency and percentage) will be used to summarize ENT/Eye examination results by treatment. In addition, the number of subjects with values of potential clinical significance determined by the investigator will be tabulated.

All ENT/Eye examination data will be listed by treatment and subject.

#### 7.10. Baseline Efficacy Evaluations

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be summarized by treatment group for the following:

Baseline average (AM/PM), AM and PM subject-reported rTNSS, iTNSS, rTOSS, iTOSS, rTNNSS and iTNNSS.

- Baseline average (AM/PM), AM and PM reflective individual nasal symptoms, instantaneous individual nasal symptoms, reflective individual non-nasal symptoms and instantaneous individual non-nasal symptoms.
- PRQLQ, PNSS.
- Individual PRQLQ scores and individual PNSS symptom scores.

#### 8. EFFICACY

The primary efficacy analysis of the primary efficacy endpoint will be performed on both the FAS (primary) and the PPS (supportive).

Table 4: Overview of Efficacy Analysis of the Primary Endpoint

| | Stats Analysis | | Stats Analysis | | Sum | mary | Individual |
|---|---|---|---|---|---|---|---|
| | Т | F | Т | F | L | | |
| Primary Endpoint: Change from Ba | seline in A | Average A | M and | PM 12- | hour rTNSS | | |
| over a 14-day Treatment Period | | | | | - 1 | | |
| Primary analysis method: (MMRM | Approac | h) | | | | | |
| rTNSS-MMRM- FAS | Y | Y | Y | | Y | | |
| rTNSS – MMRM – PPS | Y | Y | Y | 10 | Y | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TF related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TF related to summaries (i.e. descriptive statistics) of the baseline, post-treatment and change from baseline for the primary efficacy analyses method.
- Individual = Represents L related to any displays of individual subject observed raw data as well as post-baseline and change from baseline presented on the SAS dataset.

#### 8.1. General Considerations

All tests will be 2-sided and at 5% level of significance unless otherwise stated.

In addition to the analyses described below, all variables will be summarized descriptively, as appropriate.

The primary goal of the analysis of the primary endpoint will be to assess the superiority of GSP 301 NS vs placebo NS treatment comparisons for the primary endpoint rTNSS.

The primary analysis will use the FAS and a supportive analysis will be based on the PPS. The interpretation of results from statistical tests will be based on the FAS. The PPS will be used to assess the robustness of the results from the statistical tests based on the FAS.

Unless otherwise stated, 'treatment' refers to treatment group as randomized, rather than based on the actual treatment received.

#### 8.2. Statement of the Null and Alternate Hypotheses

The primary endpoint is the change from baseline in average AM and PM subject-reported 12-hour rTNSS over the 14-day treatment period.

A significance test will be made for the primary endpoint in order to assess for superiority of GSP 301 NS versus placebo NS. Demonstration of superiority for this treatment comparison will be based on a hypothesis testing approach, whereby the null hypothesis is that there is no difference between treatment groups and the alternative hypothesis is that there is a difference between the treatment groups.

A 2-sided 5% risk associated with incorrectly rejecting the null hypothesis (significance level) is considered acceptable for this study.

#### 8.3. Subgroup Analyses

The following subgroups of clinical interest will also be summarized for the FAS only, by treatment group and by day, for rTNSS: age group (6-<9, 9-<12), gender (female/male), race (American Indian or Alaska Native, Asian, Black/African American, Other and White) and ethnicity (Hispanic or Latino and Not Hispanic or Latino). iTNSS, rTOSS and PRQLQ will be analyzed only for the age subgroups (6-<9, 9-<12).

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be provided for baseline, post treatment and change from baseline.

Also, the MMRM analysis of rTNSS will be repeated for each of the age subgroups (6-<9, 9-<12).

Further subgroup analyses might be performed on an ad-hoc basis if deemed necessary.

### 8.4. Multiple Comparisons and Multiplicity

Treatment comparisons will begin with the primary endpoint. If the resulting two-sided p-value is less than 0.05, then the next comparison of the secondary endpoint will be made, in the order of clinical importance, as outlined below.

- Change from baseline in average AM and PM subject-reported 12-hour instantaneous Total Nasal Symptom Score (iTNSS) over the 14-day treatment period.
- Change from baseline in the overall Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) score on Day 15 (Visit 4) between treatment groups.
- Change from baseline in average AM and PM subject-reported 12-hour reflective Total Ocular Symptom Score (rTOSS) over the 14-day treatment period.

The testing procedure will continue until either all comparisons of interest are made, or until the point at which the resulting two-sided p-value is greater than 0.05. Once one of the tests is not significant, the testing will no longer be performed for the remainder of the endpoints.

Note: p-values for all treatment comparisons will still be displayed in the outputs of interest. The hierarchical testing will be applied when interpreting the analysis in the CSR.

No multiplicity adjustments will be made.

#### 8.5. Analysis of the Primary Efficacy Endpoint

#### 8.5.1. Primary Efficacy Analysis

The primary endpoint, change from baseline in average AM and PM subject-reported 12-hour rTNSS over a 14-day treatment period, will be evaluated using a mixed-effect repeated measures (MMRM) model. The model will adjust for study treatment, site, baseline 12-hour rTNSS and study day as the within-subject effect, with the assumption that any missing data is missing at random (MAR).

The interactions of site-by-treatment and baseline-by-treatment will be investigated separately using two independent models and will only be included in the final model if they are statistically significant at the alpha=5% level. In order to determine the interaction/s to be included in the final model, the following model-fitting process will be followed:

- 1. The main-effects model containing study treatment, site, baseline 12-hour rTNSS and study day will be fitted first:
  - a. Unstructured covariance will initially be assumed.
  - b. If the model does not converge using the unstructured covariance structure, the autoregressive (order 1) AR(1) structure will be used.
  - c. If the AR(1) structure also does not converge, other covariance structures deemed appropriate to fit the data will be used.
- 2. Two independent models will be fitted using the covariance structure of the model that converged in step 1: one model containing the site-by-treatment interaction and the other model containing the baseline-by-treatment interaction. If the interaction term is significant, it will be included in the final model. If convergence is not obtained after adding both of the interaction terms (if both are significant), the more significant interaction term will be kept in the model. Any interaction term that make model not converge will not be added to the final model.

The statements of a SAS® PROC MIXED analysis would be (if the interactions of treatment\*baseline and treatment\*site are not statistically significant):

PROC MIXED;
CLASS subject treatment site day;
MODEL change = treatment site baseline day;
REPEATED day / SUBJECT = subject TYPE=UN;
LSMEANS treatment / CL DIFF E;
ODS OUTPUT LSMEANS=Ismeans;
ODS OUTPUT DIFFS=diffs;
RUN;
QUIT;

The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-

values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be provided for baseline, post treatment and change from baseline by treatment group and day.

#### 8.6. Analysis of the Secondary Efficacy Endpoints

The secondary endpoints will be analyzed in the following order of importance (high to low):

- Change from baseline in average AM and PM subject-reported 12-hour instantaneous Total Nasal Symptom Score (iTNSS) over the 14-day treatment period.
- Change from baseline in the overall Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) score on Day 15 (Visit 4) between treatment groups.
- Change from baseline in average AM and PM subject-reported 12-hour reflective Total Ocular Symptom Score (rTOSS) over the 14-day treatment period.

Table 5 provides an overview of the planned secondary efficacy analyses.

Table 5: Overview of Planned Secondary Efficacy

| | Stats A | nalysis | Summary | | Individual |
|---|---|---|---|---|---|
| | Т | F | Т | F | L |
| Change from Baseline in Averag | e AM and | PM 12- | hour iT | NSS o | ver a 14-day |
| Treatment Period (MMRM Appr | oach) | | | | 11.55 |
| iTNSS – MMRM – FAS | Y | Y | Y | | Y |
| iTNSS – MMRM – PPS | Y | Y | Y | | |
| Change from Baseline in PRQLO | on Day | 5 (ANC | OVA | model) | |
| PRQLQ – ANCOVA – FAS | Y | Y | Y | | Y |
| Change from Baseline in Averag | e AM and | PM 12- | hour r | COSS | over a 14-day |
| Treatment Period (MMRM Appr | roach) | | | | |
| rTOSS – MMRM - FAS | Y | Y | Y | | Y |
| rTOSS – MMRM - PPS | Y | Y | Y | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TF related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TF related to summaries (i.e. descriptive statistics) of the baseline, post-treatment and change from baseline for the primary efficacy analyses method.

• Individual = Represents L related to any displays of individual subject observed raw data as well as post-baseline and change from baseline presented on the SAS dataset.

#### 8.6.1. Analysis of Change from Baseline in iTNSS and rTOSS

The analysis of change from baseline in iTNSS and rTOSS will use both the FAS (primary) and the PPS (supportive).

Similar to the primary analysis for the primary endpoint in section 8.5.1 above, the secondary endpoints (iTNSS and rTOSS) will be evaluated using a MMRM model, adjusting for covariates that include treatment, site, baseline and study day as the within-subject effect. The interactions of site-by-treatment and baseline-by-treatment will be investigated separately in the model and will only be included in final model if they are statistically significant at the alpha=5% level. An unstructured (UN) covariance will be assumed. If the model does not converge using the unstructured covariance structure, the autoregressive (order 1) AR(1) structure will be used. If this also does not converge other covariance structures deemed appropriate to fit the data will be used. The SAS® code will be similar to the primary endpoint.

The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be provided for baseline, post treatment and change from baseline by treatment group and day.

8.6.2. Analysis of Change from Baseline in the Overall PROLO on Day 15

The change from baseline in the overall PRQLQ at Day 15 (Visit 4) will be analyzed for the FAS using an ANCOVA model adjusting for study treatment, site, and baseline PRQLQ (linear, continuous covariate). The interactions of site-by-treatment and baseline PRQLQ-by-treatment group will be investigated separately in the ANCOVA model and will only be included in the final model if they are statistically significant at the alpha=5% level. Baseline is defined as the PRQLQ score at Day 1 (Visit 2). For subjects who withdrew early from the study the PRQLQ score at their discontinuation visit will be used, regardless of what actual study day this visit occurred on.

The statements of a SAS® PROC MIXED analysis would be:

proc mixed; class treatment site; model change = treatment site baseline; lsmeans treatment / cl diff; ods output lsmeans=lsmeans; ods output diffs=diffs; run; quit; The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be provided for baseline, post treatment and change from baseline by treatment group.

#### 8.7. Efficacy Analyses of Other Endpoints of Interest

The analysis on endpoints including nasal symptoms, non-nasal symptoms, individual domains of PRQLQ and PNSS will be based on the FAS. Outputs based on the PPS will be produced only on an as needed basis for these endpoints, depending on the results from the primary and secondary endpoints.

Similar methods as described for the primary endpoint above will be applied, for the other endpoints nasal symptoms, ocular symptoms and non-nasal symptoms as listed in Section 3.2.3. Similar to the primary analysis for the primary endpoint in section 8.5.1 above, these other endpoints (nasal symptoms, non-nasal symptoms and ocular symptoms) will be evaluated using a MMRM model, adjusting for covariates treatment, site, baseline and study day as the within-subject effect. The interaction term day-by-treatment will also be included in the MMRM model for the by-day analysis for rTNSS and iTNSS. The individual symptom analysis will be conducted by including a 'by individual symptom' statement to the proc mixed model. An unstructured (UN) covariance will be assumed. If the model does not converge using the UN covariance structure, the autoregressive-order 1 (AR(1)) structure will be used. If this also does not converge other covariance structures deemed appropriate to fit the data will be used. The SAS® code will be similar to the primary endpoint. If there is no convergence for the MMRM model with day-by-treatment term, ANCOVA model will be used to present the by-day estimates for rTNSS and iTNSS.

Similar to the analysis for the secondary endpoint in Section 8.6.2 above, the other endpoints overall PNSS and individual domains PNSS, PRQLQ will be evaluated using an analysis of covariance (ANCOVA) model adjusting for covariates that include treatment, site and baseline. The individual domain analysis will be conducted by including a 'by individual domain' statement to the proc mixed model.

The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. For some of the endpoints the adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals. For the by-day analysis, the above will be presented for each day. For the individual symptom/domain analysis, the above will be presented for each symptom/domain.

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be provided for baseline, post treatment and change from baseline by treatment group (and by day for certain endpoints) for each endpoint detailed above.

# 8.8. Summary of Reasons for Efficacy Non-Evaluability/Exclusion from Efficacy Analyses

The reasons for excluding subjects from the PPS will be listed by treatment and subject.

#### 9. SAFETY AND TOLERABILITY

#### 9.1. Overall Summary of Tolerability

The safety analyses will be based on the SAS, unless otherwise specified. If a subject is randomized in the study more than one time, it will be decided at the Blind Data Review Meeting (BDRM) or after unblinding, on a case by case basis if the subject is counted in the numerator of any specific safety analysis.

Table 6 provides an overview of the planned analyses.

Table 6: Overview of Planned Safety Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Adverse Events | | | |
| Overview | Y[2] | | |
| Treatment Emergent AEs | Y[1][2] | | Y |
| Treatment Emergent AEs Severity | Y[2] | | Y |
| Treatment-Related Emergent AEs | Y[2] | | Y |
| Placebo Run-In Period AEs | Y[2] | | Y |
| Pre-run-in period AEs | | | Y |
| AEs Leading to Withdrawal | | | Y |
| SAEs | Y[2] | | Y |
| Treatment Emergent SAEs | Y[2] | | Y |
| Treatment Emergent SAEs Severity | Y[2] | | Y |
| Treatment-Related Emergent SAEs | Y[2] | | |
| Laboratory | 1 | | |
| Pregnancy Test Results | | | Y |
| Other | | 11 - 11 11 | |
| Vital Signs | Y[3] [2] | | Y |
| Physical Examination | Y[4] [2] | | Y |
| Focused ENT Examination | Y[5] [2] | | Y |

#### NOTES:

- Y = Yes display generated.
- [1]: Display will also be produced by SOC, severity, and by relationship to study medication
- [2]: Display will be based on safety analysis set
- [3]: Display will be produced separately for overall summary (inc. change from baseline), for potentially clinically significant results, and shift tables
- [4]: Display will be produced separately for overall summary
- [5]: Display will be produced separately for overall summary and for potentially clinically significant results

# 9.2. Adverse Event Preferred Term and Body/Organ System Summary Tables

#### 9.2.1. Summaries of Adverse Event Incidence Rates for All Subjects

Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 21.0.

All AEs will be displayed in listings.

Any AE that occurs during the placebo run-in period will be summarized separately from the AEs occurring during the randomized treatment period. Any AE that occurs pre-run-in (between the subjects signing informed consent and administration of the first dose of the run-in study medication) will be listed. Adverse events occurring after the first dose of the randomized study medication will be defined as treatment-emergent adverse events (TEAEs).

A comparison of the incidence rate of AEs between study treatment groups will be presented overall, occurring in greater or equal to 1%, 2%, 3%, as well as AEs occurring in the study treatment arm in higher frequency than in placebo arm. Incidence rate is determined by the number of subjects with AEs divided by the total duration (day) of treatment across all subjects in given treatment group, multiplied by 100.

Summaries of the number of subjects with TEAEs and the number of TEAEs experienced will be presented by treatment. The number of subjects and the number of TEAEs will be presented using frequency counts and percentages, overall and by system organ class (SOC) and preferred term (PT). The percentages will be calculated as the number of subjects with TEAEs divided by the number of subjects in each treatment in the safety analysis set. Tables of the number and percentage of subjects and the number of TEAEs by intensity and by relationship to study medication will also be presented. If severity of an event is missing, then set AE severity as "Severe". If relationship to study treatment is missing, then set relationship as "Related". Similar tables will be created for treatment related emergent AEs (TREAEs). Events will be assigned to the study treatment administered prior to the start of the TEAE. Events that occurred during discharge and final follow-up will be assigned to the study treatment administered prior to the start of the event.

#### 9.2.2. Missing and Partial AE Dates

Due diligence will be done to obtain accurate AE information. If all planned methods to obtain accurate AE information have failed, missing and partial AE onset and end dates will be imputed. Imputed dates will be flagged in the individual supportive subject listings. Unless otherwise specified, the following conventions will be used:

Missing and Partial AE onset dates

- If onset date is completely missing, then onset date is set to date of first dose
- If onset year is present and
  - o month and day are missing:
    - If onset year = year of first dose, then set onset date to date of first dose

- If onset year < year of first dose, then set onset month and day to December 31st.
- If onset year > year of first dose, then set onset month and day to January
   1st
- o month is missing:
  - If onset year = year of first dose, then set onset date to date of first dose
  - If onset year < year of first dose, then set onset month to December
  - If onset year > year of first dose, then set onset month to January
- If onset month and year are present and day is missing:
  - o If onset year = year of first dose and
    - onset month = month of first dose then set onset date to date of first dose
    - onset month < month of first dose then set onset date to last day of month
    - onset month > month of first dose then set onset date to 1st day of month
  - o If onset year < year of first dose then set onset date to last day of month
  - o If onset year > year of first dose then set onset date to 1st day of month
- For all other cases, set onset date to date of first dose

#### Missing and Partial AE end dates

- If end date is completely missing, end date is not imputed and the AE is flagged as "ongoing"
- If year is present and
  - o month and day are missing
    - If year = year of last dose, then set end date to the date of last dose
    - If year < year of last dose, then set end month and day to December 31st</p>
    - If year > year of last dose, then set end month and day to January 1st
  - o month is missing
    - If year = year of last dose, then set end date to date of last dose
    - If year < year of last dose, then set end month to December</p>
    - If year > year of last dose, then set end month to January
- If month and year are present and day is missing:
  - o If year = year of last dose and
    - month = month of last dose then set day to day of last dose
    - month < month of last dose then set day to last day of month

- month > month of last dose then set day to 1st day of month
- o If year < year of last dose, then set end date to last day of the month
- o If year > year of last dose, then set end date to 1st day of month
- For all other cases, set end date to date of last dose

# 9.2.3. Summaries of Adverse Incidence Rates for Serious Adverse Events (SAE), adverse events leading to discontinuation, and treatment-related emergent adverse events

The number and percentage of TEAEs, SAEs, AEs leading to discontinuation, treatment-related emergent AEs and treatment-related emergent SAEs will be summarized by SOC, PT, and treatment group. The percentages will be calculated as the number of subjects with AEs divided by the number of subjects in each treatment in the safety analysis set. Tables of the number and percentage of subjects and the number of AEs by intensity and by relationship to study medication will also be presented.

Any withdrawals will be listed and summarized by reason for withdrawal, treatment and by any other relevant categorical information.

# 9.3. Total Duration of Therapy, treatment Compliance and diary compliance

The number of subjects exposed to each study treatment will be summarized.

The number of days on treatment and the number of days on study (including run-in period and treatment periods) will be summarized by study treatment.

Treatment compliance will be calculated (the total number of doses actually taken / total number of doses expected\*100). For subjects who have completed the study:

| | | Compliance Criteria | | |
|---|---|---|---|---|
| Study<br>Period | Duration | Scheduled<br>Doses | Not more than 125% (doses) | Not less<br>than 75%<br>(doses) |
| Randomized<br>Treatment | 14 Days | 28 | 35 | 21 |

For subjects who are early terminated, treatment compliance will be determined from their duration on treatment, up to the time they are considered completed or early terminated. If a patient is on randomized treatment for more than 14 days, use 14 as denominator to determine treatment compliance. Subjects taking fewer than 75% or more than 125% of the required doses will be considered non-compliant with dosing.

In addition, treatment compliance will be classified into four categories (<75%, >=75% - <=100%, >100% - =<125%, >125%). Treatment compliance will be summarized by category and study treatment.

Diary compliance (number of diary entry missed by visit) will only be presented in the listing.

#### 9.4. Concomitant and Other Medications

At Visit 1 subjects will be questioned about current concomitant medication use. At Visit 2, Visit 3 and Visit 4 subjects will be questioned about ongoing or new concomitant medication use.

Concomitant medications are defined as medications either ongoing or ended on or after the first dose of study medication. All concomitant medications taken since screening until the end of the study will be listed by treatment and subject. If the end date and 'ongoing' are missing, then the medication will be considered as concomitant medication. Medication taken after last randomized treatment will be identified and flagged in the listing.

#### 9.4.1. Missing and Partial Concomitant and Other Medication Start and Stop Dates

For the purpose of inclusion in prior and/or concomitant medication tables, incomplete medication start and stop dates will be imputed as follows:

- If year and month are present and day is missing, then set day to first day of month for start date, and set day to last day of month for end date
- If year and day are present and month is missing, then set month to January for start date, and set month to December for end date
- If year is present and month and day are missing, then set month and day to January 1 for start date, and set month and day to December 31 for end date
- Completely missing date will not be imputed

The partial dates will be provided as such in the subject data listings (with the imputed dates).

#### 9.5. Pregnancy Test

All females of child bearing potential will have a urine pregnancy test at Visits 1, 2 and final Visit 4.

Pregnancy test results will be listed by treatment and subject.

#### 9.6. Vital Signs

The subject's post-baseline vital signs will be recorded (pulse rates, sitting systolic and diastolic blood pressure) at Visits 3 and 4. Height and weight will also be recorded at Visit 4. Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be used to summarize vital sign results and changes from baseline by treatment group and visit.

Values outside the respective normal range and values deemed as clinically significant by the Investigator will be listed. Normal ranges for pulse rate, systolic BP and diastolic BP are listed in Table 7.

Table 7: Normal ranges of vital signs <sup>6,7</sup>

| Vital Sign | Abnormal Criteria |
|---|---|
| Pulse Rate (Beats/min) | Pulse rate: 6-11 years and Result is <60 or >95 |
| Systolic BP (mmHG) | Systolic BP: 6-9 years and Result is <95 or >110 Systolic BP: 10-11 years and Result is <100 or >119 |
| Diastolic BP(mmHG) | Diastolic BP: 6-9 years and Result is <60 or >73 Diastolic BP: 10-11 years and Result is <65 or >76 |

The number of subjects with values of potential clinical significance determined by the investigator will be tabulated by treatment group and visit.

All vital sign data will be listed by treatment and subject.

#### 9.7. Physical Examination

Post-baseline physical examinations (comprehensive) will be performed at the Final Visit (Visit 4).

Descriptive statistics (frequency and percentage) will be used to summarize physical examination results by body system, treatment group and visit. In addition, the number of subjects with values of potential clinical significance determined by the investigator will be tabulated.

All physical examination data will be listed by treatment and subject.

#### 9.8. Focused ENT/Eye examination

Post-baseline focused ENT/Eye examinations will be performed at Visits 3 and 4.

Descriptive statistics (frequency and percentage) will be used to summarize ENT/Eye examination results by treatment group and visit. In addition, the number of subjects with values of potential clinical significance determined by the investigator will be tabulated.

The focused ENT exam reviews the following 9 symptoms: Nasal irritation, Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal Erythema, Crusting of Mucosa, Throat Irritation, Candidiasis, Post Nasal Drip. A severity grade of "None" is collected on the CRF and considered as a normal value; more severe grades are considered as abnormal value.

For eye examination, results of both left and right eye are considered. The overall evaluation for each subject is determined by the more severe result from either one of the eyes.

All ENT/Eye examination data will be listed by treatment and subject.

#### 9.9. Study Termination Status

A subject may voluntarily discontinue study participation at any time after giving informed consent and before the completion of the last visit of the study. The Investigator may also discontinue the subject's study participation at any time at his/her discretion and for any reason.

The reasons for subject withdrawal will be recorded and may include, but are not limited to:

- 1. Withdrawal of consent by the subject to continue in the study.
- 2. Development of a serious or intolerable AE that necessitates discontinuation at the discretion of the Investigator (AE section of the case report form/electronic case report form [CRF/eCRF] must be completed; includes serious adverse event [SAE], death).
- 3. At the discretion of the Investigator, when he/she believes continued participation is not in the best interest of the subject.
- 4. At the discretion of the Investigator, when the subject does not adhere to the study procedures.
- 5. A protocol deviation that, in the opinion of the Sponsor and the Investigator, warrants discontinuation from the study.

On leaving the study, either at the scheduled end of treatment and subsequent follow-up, or following early withdrawal from the study, or at such time when the patient is considered to be lost to follow-up, the date and reason for leaving the study will be recorded.

If there are multiple reasons for early withdrawal/discontinuation, the worst-case scenario should be chosen. Early discontinuation data will be listed by treatment and subject. Early discontinuations due to Inclusion/Exclusion (I/E) criteria violation, in SAS subjects, will be summarized by treatment and I/E criteria.

December 06, 2018

## 10. CHANGES IN ANALYSES FROM THE PROTOCOL

None

#### 11. REFERENCES

- Allergic Rhinitis: Developing Drug Products for Treatment. Guidance for Industry (Draft Guidance); February 2016, <a href="http://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm071293.pdf">http://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm071293.pdf</a>.
- 2. Barnes ML, Vaidyanathan S, Williamson PA, Lipworth BJ. The minimal clinically important difference in allergic rhinitis. Clin Exp Allergy. 2010;40(2):242-250.
- 3. Juniper EF and Guyatt HG. Development and testing of a new measure of health status for clinical trials in rhinoconjunctivitis. Clin and Experimental Allergy 1991;21:77-83.
- 4. US Prescribing Information: DYMISTA (azelastine hydrochloride and fluticasone propionate) Nasal Spray; Initial U.S. Approval: 2012.
- 5. Meltzer EO, Schatz M, Nathan R, Garris C, Stanford RH, Kosinski M. Reliability, validity, and responsiveness of the rhinitis control assessment test in patients with rhinitis. J Allergy Clin Immunol 2013;131:379-386.
- 6. Kliegman, RM, Stanton BMD, Geme JS, Schor NF. Nelson Textbook of Pediatrics, 20th Edition. Philadelphia, PA: Elsevier.
- 7. Weaver DJ. "Hypertension in Children and Adolescents." Pediatrics in Review 38.8 August 2017: 369-382.

# List of Tables

| Section 14.1 - Demographic, baseline and other subject-specific characteristics |
|---|
| Table 14.1.1 Summary of Subject Disposition (All Subjects) |
| Table 14.1.2.1 Summary of Protocol Deviations during Pre-run-in Period (All Enrolled Subjects) |
| Table 14.1.2.2 Summary of Protocol Deviations during Placebo Run-In Period (Run-in Set) |
| Table 14.1.2.3 Summary of Protocol Deviations during Randomized Treatment Period (Safety Analysis Set) |
| Table 14.1.2.4 Summary of Major Protocol Deviations (Safety Analysis Set)72 |
| Table 14.1.3.1 Summary of Analysis Populations |
| Table 14.1.4.1 Summary of Demographic Data (Run-in Set) |
| Table 14.1.4.2 Summary of Demographic Data (Safety Analysis Set)76 |
| Table 14.1.4.3 Summary of Demographic Data (Full Analysis Set)77 |
| Table 14.1.4.4 Summary of Demographic Data (Per Protocol Set)77 |
| Section 14.2.1 Primary endpoint rTNSS |
| Table 14.2.1.1 Summary of Average AM and PM rTNSS by Day (Full Analysis Set)78 |
| Table 14.2.1.2 Summary of Repeated Measures Analysis Results of Average AM and PM rTNSS over the 14-day Treatment Period (Full Analysis Set)79 |
| Table 14.2.1.3 Summary of Average AM and PM rTNSS by Day (Per Protocol Set)80 |
| Table 14.2.1.4 Summary of Repeated Measures Analysis Results of Average AM and PM rTNSS over the 14-day Treatment Period (Per Protocol Set)80 |
| Table 14.2.1.5 Subgroup Analyses (Age Group): Summary of Average AM and PM rTNSS by Day (Full Analysis Set) |
| Table 14.2.1.6 Subgroup Analyses (Age Group): Summary of Repeated Measures Analysis Results of Average AM and PM rTNSS over the 14-day Treatment Period (Full Analysis Set) |
| Table 14.2.1.7 Subgroup Analyses (Sex): Summary of Average AM and PM rTNSS by Day (Full Analysis Set) |

| Table 14.2.1.8 Subgroup Analyses (Race): Summary of Average AM and PM rTNSS by Day (Full Analysis Set)8 | 4 |
|---|---|
| Table 14.2.1.9 Subgroup Analyses (Ethnicity): Summary of Average AM and PM rTNSS by Day (Full Analysis Set) | 5 |
| Section 14.2.2 Secondary endpoints iTNSS, rTOSS and PROLQ | |
| Table 14.2.2.1.1 Summary of Average AM and PM iTNSS by Day (Full Analysis Set)8 | 6 |
| Table 14.2.2.1.2 Summary of Repeated Measures Analysis Results of Average AM and PM iTNSS over the 14-day Treatment Period (Full Analysis Set)8 | 6 |
| Table 14.2.2.1.3 Summary of Average AM and PM iTNSS by Day (Per Protocol Set)8 | 6 |
| Table 14.2.2.1.4 Summary of Repeated Measures Analysis Results of Average AM and PM iTNSS over the 14-day Treatment Period (Per Protocol Set)8 | 6 |
| Table 14.2.2.1.5 Subgroup Analyses (Age Group): Summary of Average AM and PM iTNSS by Day (Full Analysis Set)8 | 6 |
| Table 14.2.2.2.1 Summary of Average AM and PM rTOSS by Day (Full Analysis Set)8 | 7 |
| Table 14.2.2.2.2 Summary of Repeated Measures Analysis Results of Average AM and PM rTOSS over the 14-day Treatment Period (Full Analysis Set)8 | 7 |
| Table 14.2.2.2.3 Summary of Average AM and PM rTOSS by Day (Per Protocol Set) | 7 |
| Table 14.2.2.2.4 Summary of Repeated Measures Analysis Results of Average AM and PM rTOSS over the 14-day Treatment Period (Per Protocol Set)8 | :7 |
| Table 14.2.2.2.5 Subgroup Analyses (Age Group): Summary of Average AM and PM rTOSS by Day (Full Analysis Set)8 | 17 |
| Table 14.2.2.3.1 Summary of the Overall PRQLQ Score and Individual Domains on Day 15 (Full Analysis Set) | 88 |
| Table 14.2.2.3.2 Summary of ANCOVA Analysis Results of the Overall PRQLQ Score and Individual Domains on Day 15 (Full Analysis Set) | 39 |
| Table 14.2.2.3.3 Subgroup Analysis (Age Group): Summary of the Overall PRQLQ Score and Individual Domains on Day 15 (Full Analysis Set)9 | 0( |
| Section 14.2.3 Other efficacy endpoints | |
| Table 14.2.3.1.1 Summary of AM rTNSS by Day (Full Analysis Set)9 | 1 |
| Table 14.2.3.1.2 Summary of Repeated Measures Analysis Results of AM rTNSS over the 14-day Treatment Period (Full Analysis Set) | )2 |
| Table 14.2.3.2.1 Summary of PM rTNSS by Day (Full Analysis Set)9 | )3 |
| Table 14.2.3.2.2 Summary of Repeated Measures Analysis Results of PM rTNSS over the 14-day Treatment Period (Full Analysis Set) | )3 |

| Table 14.2.3.3.1 Summary of AM iTNSS by Day (Full Analysis Set) | 93 |
|---|---|
| Table 14.2.3.3.2 Summary of Repeated Measures Analysis Results of AM iTNSS over the 14-day Treatment Period (Full Analysis Set) | 94 |
| Table 14.2.3.4.1 Summary of PM iTNSS by Day (Full Analysis Set) | 94 |
| Table 14.2.3.4.2 Summary of Repeated Measures Analysis Results of PM iTNSS over the 14-day Treatment Period (Full Analysis Set) | 94 |
| Table 14.2.3.5.1 Summary of Average AM and PM Reflective Individual Nasal Symptoms by Day (Full Analysis Set) | 95 |
| Table 14.2.3.5.2 Summary of Repeated Measures Analysis Results of Average AM and PM Reflective Individual Nasal Symptoms over the 14-day Treatment | 96 |
| Table 14.2.3.6.1 Summary of AM Reflective Individual Nasal Symptoms by Day (Full Analysis Set) | 97 |
| Table 14.2.3.6.2 Summary of Repeated Measures Analysis Results of AM Reflective Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set) | 97 |
| Table 14.2.3.7.1 Summary of PM Reflective Individual Nasal Symptoms by Day (Full Analysis Set) | 97 |
| Table 14.2.3.7.2 Summary of Repeated Measures Analysis Results of PM Reflective Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set) | 97 |
| Table 14.2.3.8.1 Summary of Average AM and PM Instantaneous Individual Nasal Symptoms by Day (Full Analysis Set) | 98 |
| Table 14.2.3.8.2 Summary of Repeated Measures Analysis Results of Average AM and PM Instantaneous Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set) | 98 |
| Table 14.2.3.9.1 Summary of AM Instantaneous Individual Nasal Symptoms by Day (Full Analysis Set) | 98 |
| Table 14.2.3.9.2 Summary of Repeated Measures Analysis Results of AM Instantaneous Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set) | 98 |
| Table 14.2.3.10.1 Summary of PM Instantaneous Individual Nasal Symptoms by Day (Full Analysis Set) | 98 |
| Table 14.2.3.10.2 Summary of Repeated Measures Analysis Results of PM Instantaneous Individual Nasal Symptoms over the 14-day Treatment Period (Full | 98 |
| Table 14.2.3.11.1 Summary of Average AM and PM iTOSS by Day (Full Analysis Set) | 99 |

| Table : | 14.2.3.11.2 Summary of Repeated Measures Analysis Results of Average AM and | |
|---|---|---|
| 14010 | PM iTOSS over the 14-day Treatment Period (Full Analysis Set) | 99 |
| Table | 14.2.3.12.1 Summary of AM rTOSS by Day (Full Analysis Set) | 99 |
| Table 1 | 14.2.3.12.2 Summary of Repeated Measures Analysis Results of AM rTOSS over the 14-day Treatment Period (Full Analysis Set) | 99 |
| Table 1 | 14.2.3.13 1 Summary of PM rTOSS by Day (Full Analysis Set) | 99 |
| Table 1 | 14.2.3.13 2 Summary of Repeated Measures Analysis Results of PM rTOSS over the 14-day Treatment Period (Full Analysis Set) | 99 |
| Table | 14.2.3.14.1 Summary of AM iTOSS by Day (Full Analysis Set) | 99 |
| Table 1 | 14.2.3.14.2 Summary of Repeated Measures Analysis Results of AM iTOSS over the 14-day Treatment Period (Full Analysis Set) | 99 |
| Table 1 | 14.2.3.15.1 Summary of PM iTOSS by Day (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.15.2 Summary of Repeated Measures Analysis Results of PM iTOSS over the 14-day Treatment Period (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.16.1 Summary of Average AM and PM rTNNSS by Day (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.16.2 Summary of Repeated Measures Analysis Results of Average AM and PM rTNNSS over the 14-day Treatment Period (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.17.1 Summary of Average AM and PM iTNNSS by Day (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.17.2 Summary of Repeated Measures Analysis Results of Average AM and PM iTNNSS over the 14-day Treatment Period (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.18.1 Summary of AM rTNNSS by Day (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.18.2 Summary of Repeated Measures Analysis Results of AM rTNNSS over the 14-day Treatment Period (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.19.1 Summary of PM rTNNSS by Day (Full Analysis Set) | 100 |
| Table 1 | 14.2.3.19.2 Summary of Repeated Measures Analysis Results of PM rTNNSS over the 14-day Treatment Period (Full Analysis Set) | 101 |
| Table 1 | 14.2.3.20.1 Summary of AM iTNNSS by Day (Full Analysis Set) | 101 |
| Table 1 | 14.2.3.20.2 Summary of Repeated Measures Analysis Results of AM iTNNSS over the 14-day Treatment Period (Full Analysis Set) | 101 |
| Table 1 | 14.2.3.21.1 Summary of PM iTNNSS by Day (Full Analysis Set) | 102 |
| Table 1 | 14.2.3.21.2 Summary of Repeated Measures Analysis Results of PM iTNNSS over the 14-day Treatment Period (Full Analysis Set) | 102 |

| Table 14.2.3.22.1 Summary of Average AM and PM Reflective Individual Non-nasal symptoms by Day (Full Analysis Set) | 102 |
|---|---|
| Table 14.2.3.22.2 Summary of Repeated Measures Analysis Results of Average AM and PM Reflective Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set) | 102 |
| Table 14.2.3.23.1 Summary of AM Reflective Individual Non-nasal symptoms by Day (Full Analysis Set) | 102 |
| Table 14.2.3.23.2 Summary of Repeated Measures Analysis Results of AM Reflective Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set) | 102 |
| Table 14.2.3.24.1 Summary of PM Reflective Individual Non-nasal symptoms by Day (Full Analysis Set) | 103 |
| Table 14.2.3.24.2 Summary of Repeated Measures Analysis Results of PM Reflective Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set) | 103 |
| Table 14.2.3.25.1 Summary of Average AM and PM instantaneous Individual Non-nasal symptoms by Day (Full Analysis Set) | 103 |
| Table 14.2.3.25.2 Summary of Repeated Measures Analysis Results of Average AM and PM instantaneous Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set) | 103 |
| Table 14.2.3.26.1 Summary of AM instantaneous Individual Non-nasal symptoms by Day (Full Analysis Set) | 103 |
| Table 14.2.3.26.2 Summary of Repeated Measures Analysis Results of AM instantaneous Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set) | 103 |
| Table 14.2.3.27.1 Summary of PM instantaneous Individual Non-nasal symptoms by Day (Full Analysis Set) | 104 |
| Table 14.2.3.27.2 Summary of Repeated Measures Analysis Results of PM instantaneous Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set) | 104 |
| Table 14.2.3.28.1 Summary of Physician Assessed Nasal Symptoms Score (PNSS) and Individual Assessments at Day 15 (Full Analysis Set) | 105 |
| Table 14.2.3.28.2 Summary of ANCOVA Analysis Results of Physician Assessment of Nasal Symptoms Score (PNSS) and individual assessments at Day 15 (Full Analysis Set) | 106 |

| 14.5.2 Mayerse event | 14.3.2 A | Adverse | event |
|----------------------|----------|---------|-------|
|----------------------|----------|---------|-------|

| 14.5.2 Adverse event | |
|---|---|
| Table 14.3.1.1 Overall Summary of Treatment Emergent Adverse Event (TEAE) (Safety Analysis Set) | 107 |
| Table 14.3.1.2 Summary of Treatment-Emergent Adverse Events (Safety Analysis Set) | 109 |
| Table 14.3.1.3 Summary of Treatment-Related Emergent Adverse Events (Safety Analysis Set) | 110 |
| Table 14.3.1.4 Summary of Treatment-Emergent Adverse Events Leading to Discontinuation (Safety Analysis Set) | 110 |
| Table 14.3.1.5 Summary of Treatment-Emergent Adverse Events by Severity (Safety Analysis Set) | 111 |
| Table 14.3.1. 6 Summary of Treatment-Emergent Adverse Events by Relationship to Study Treatment (Safety Analysis Set) | 112 |
| Table 14.3.1. 7 Summary of Treatment-Emergent Serious Adverse Events (Safety Analysis Set) | 113 |
| Table 14.3.1. 8 Summary of Treatment- Emergent Related Serious Adverse Events (Safety Analysis Set) | 113 |
| Table 14.3.1.9 Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Analysis Set) | 113 |
| Table 14.3.1. 10 Summary of Treatment-Related Emergent Adverse Events (TEAE) Leading to Discontinuation of the Study (Safety Analysis Set) | 113 |
| Table 14.3.1. 11 Summary of Treatment-Emergent Adverse Events with frequency >= 1% (Safety Analysis Set) | 113 |
| Table 14.3.1. 12 Summary of Treatment-Emergent Adverse Events with frequency >= 2% (Safety Analysis Set) | 113 |
| Table 14.3.1. 13 Summary of Treatment-Emergent Adverse Events with frequency >= 3% (Safety Analysis Set) | 113 |
| Table 14.3.1. 14 Summary of Treatment-Emergent Adverse Events with frequency higher in GSP 301 NS group than in Placebo NS group (Safety Analysis Set) | 113 |
| Table 14.3.1. 15 Overall Summary of Adverse Events during Placebo Run-in Period (Run-in Set) | 113 |
| Table 14.3.1. 16 Overall Summary of Adverse Events Pre-run-in (All Subjects) | 114 |
| 14.3.2 Vital Signs, Physical Exam, focused ENT/Eye Results and exposure | |
| Table 14.3.2.1.1 Summary of Vital Signs (Safety Analysis Set) | 115 |
| Table 14.3.2.1.2 Summary of Potentially Clinically Significant Vital Signs (Safety Analysis Set) | 117 |

| Glenmark Specialty S.A. |
|----------------------------|
| Statistical Analysis Plan |
| Study Number - GSP 301-305 |

## December 06, 2018

| Table 14.3.2.2.1 | Summary of Physical Examination (Safety Analysis Set) | 118 |
|---|---|---|
| Table 14.3.2.3.1 | Summary of Focused ENT Examination (Safety Analysis Set) | 119 |
| | 2 Summary of Potentially Clinical Significant Focused ENT Examination fety Analysis Set) | 120 |
| | Summary of Potentially Clinical Significant Eye Examination (Safety alysis Set) | 121 |
| | Summary of Extent of Exposure during the Randomized Treatment od (Safety Analysis Set) | 122 |

# **List of Listings**

| Section 16.1 - Demographic, baseline, concomitant meds, medical history and other subject-specific characteristics | |
|---|---|
| Listing 16.2.1.1 Listing of Eligibility | 123 |
| Listing 16.2.1.2 Listing of Discontinued Subjects (All Subjects) | 124 |
| Listing 16.2.2.1 Listing of Protocol Deviations (All Subjects) | 125 |
| Listing 16.2.3.1 Listing of Subjects Excluded from the Full Analysis Set (Safety Analysis Set) | 126 |
| Listing 16.2.3.2 Listing of Subjects Excluded from the Per Protocol Set (Safety Analysis Set) | 127 |
| Listing 16.2.4.1 Listing of Demographics (Safety Analysis Set) | 128 |
| Listing 16.2.4.2 Listing of Medical History (Safety Analysis Set) | 129 |
| Listing 16.2.4.3 Listing of Prior and Concomitant Medications (Safety Analysis Set) | 130 |
| Listing 16.2.4.4 Listing of Skin Prick Test/Allergy Testing (Safety Analysis Set) | 132 |
| Listing 16.2.4.5 Listing of Pollen Counts and Rainfall by Site (Safety Analysis Set) | 133 |
| Listing 16.2.4.6 Listing of Subject Visits (Safety Analysis Set) | 134 |
| Listing 16.2.5.1 Listing of Drug Accountability (Safety Analysis Set) | 135 |
| Listing 16.2.5.2 Listing of Treatment and Dairy Compliance (Safety Analysis Set) | 136 |
| Listing 16.2.5.3 Listing of Extent of Exposure (Safety Analysis Set) | 137 |
| Section 16.2 – Efficacy | |
| Listing 16.2.6.1 Listing of AM and PM Allergic Rhinitis Symptom Evaluation (Reflective Nasal Symptom Scores) (Safety Analysis Set) | 138 |
| Listing 16.2.6.2 Listing of AM and PM Allergic Rhinitis Symptom Evaluation (Instantaneous Nasal Symptom Scores) (Safety Analysis Set) | 139 |
| Listing 16.2.6.3 Listing of Subject-reported AM, PM and average AM and PM rTNSS (Safety Analysis Set) | 140 |
| Listing 16.2.6.4 Listing of Subject-reported AM, PM and average AM and PM iTNSS (Safety Analysis Set) | 141 |
| Listing 16.2.6.5 Listing of AM and PM Reflective Non-Nasal Symptom Scores (Safety Analysis Set) | 142 |
| Listing 16.2.6.6 Listing of AM and PM Instantaneous Non-Nasal Symptom Scores (Safety Analysis Set) | 143 |

| Listing 16.2.6.7 Listing of Subject-reported AM, PM and average AM and PM rTNNSS (Safety Analysis Set) | 144 |
|---|---|
| Listing 16.2.6.8 Listing of Subject-reported AM, PM and average AM and PM iTNNSS (Safety Analysis Set) | 145 |
| Listing 16.2.6.9 Listing of Subject-reported AM, PM and average AM and PM rTOSS (Safety Analysis Set) | 146 |
| Listing 16.2.6.10 Listing of Subject-reported AM, PM and average AM and PM iTOSS (Safety Analysis Set) | 147 |
| Listing 16.2.6.11 Listing of Pediatric Rhinoconjunctivitis Quality of Life (PRQLQ) (Safety Analysis Set) | 148 |
| Listing 16.2.6.12 Listing of Physician Assessed Nasal Symptom Scores (PNSS) (Safety Analysis Set) | 149 |
| Section 16.3 – Safety | |
| Listing 16.2.7.1 Listing of Treatment Emergent Adverse Events by Treatment During Randomized Treatment Period (Safety Analysis Set) | 150 |
| Listing 16.2.7.2 Listing of Adverse Events During Placebo Run-in Period (Run-in Set) | 151 |
| Listing 16.2.7.3 Listing of Adverse Events During Pre-run-in Period (All Subjects) | 151 |
| Listing 16.2.7.4 Listing of Adverse Events Leading to Withdrawal (All Subjects) | 151 |
| Listing 16.2.7.5 Listing of Serious Adverse Event During Randomized Treatment Period (Safety Analysis Set) | 151 |
| Listing 16.2.7.6 Listing of Serious Adverse Event During Placebo Run-in Period (Run-in Set) | 151 |
| Listing 16.2.7.7 Listing of Serious Adverse Event During Pre-run-in Period (All Subjects) | 151 |
| Listing 16.2.7.8 Listing of of Death (All Subjects) | 152 |
| Listing 16.2.8.1 Listing of Pregnancy Test Results (Safety Analysis Set) | 153 |
| Listing 16.2.8.2 Listing of Physical Examination (Safety Analysis Set) | 154 |
| Listing 16.2.8.3 Listing of Focused ENT Examination (Safety Analysis Set) | 155 |
| Listing 16.2.8.4 Listing of Eye Examination (Safety Analysis Set) | 156 |
| Listing 16.2.8.5 Listing of Vital Signs (Safety Analysis Set) | 157 |

#### List of Figures

- Figure 11.2.1.1.1 LS Means with 95% Cls of Change in Average AM and PM rTNSS Over the 14-day Treatment Period (Full Analysis Set)
- Figure 11.2.1.1.2 LS Means with 95% Cls of Change in average AM and PM rTNSS Over the 14-day Treatment Period (Per Protocol Set)
- Figure 11.2.1.2.1 LS Means with 95% CIs of Change in average AM and PM iTNSS Over the 14-day Treatment Period (Full analysis Set)
- Figure 11.2.1.2.2 LS Means with 95% CIs of Change in average AM and PM iTNSS Over the 14-day Treatment Period (Per Protocol Set)
- Figure 11.2.1.3.1 LS Means with 95% CIs of Change in average AM and PM rTOSS Over the 14-day Treatment Period (Full analysis Set)
- Figure 11.2.1.3.2 LS Means with 95% CIs of Change in average AM and PM rTOSS Over the 14-day Treatment Period (Per Protocol Set)
- Figure 11.2.1.4 LS Means with 95% CIs of Change in PRQLQ Score from Baseline to Day 15 (Full Analysis Set)
- Figure 11.2.1.5 LS Means with 95% CIs of Change in average AM and PM iTOSS Over the 14-day Treatment Period (Full Analysis Set)
- Figure 11.2.1.6 LS Means with 95% CIs of Change in average AM and PM rTNNSS Over the 14-day Treatment Period (Full Analysis Set)
- Figure 11.2.1.7 LS Means with 95% CIs of Change in average AM and PM iTNNSS Over the 14-day Treatment Period (Full Analysis Set)
- Figure 11.2.1.8.1 Treatment Differences of LS Means with 95% CIs of Average AM and PM rTNSS Over the 14-day Treatment Period (Full Analysis Set)
- Figure 11.2.1.8.2 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM rTNSS Over the 14-day Treatment Period (Per Protocol Set)
- Figure 11.2.1.9.1 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM iTNSS Over the 14-day Treatment Period (Full analysis Set)
- Figure 11.2.1.9.2 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM iTNSS Over the 14-day Treatment Period (Per Protocol Set)
- Figure 11.2.1.10.1 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM rTOSS Over the 14-day Treatment Period (Full analysis Set)
- Figure 11.2.1.10.2 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM rTOSS Over the 14-day Treatment Period (Per Protocol Set)
- Figure 11.2.1.11 Treatment Differences of LS Means with 95% CIs of Change in PRQLQ Score from Baseline to Day 15 (Full Analysis Set)

Figure 11.2.1.12 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM iTOSS Over the 14-day Treatment Period (Full Analysis Set)

Figure 11.2.1.13 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM rTNNSS Over the 14-day Treatment Period (Full Analysis Set)

Figure 11.2.1.14 Treatment Differences of LS Means with 95% CIs of Change in average AM and PM iTNNSS Over the 14-day Treatment Period (Full Analysis Set)

Table 14.1.1 Summary of Subject Disposition (All Subjects)

| | | Number (%) of subjects | |
|---|---|---|---|
| · | Placebo NS | GSP 301 NS | Total |
| Subjects | (N=xxx) | (N=xxx) | (N=xxx) |
| Total screened | | | XXX |
| Screen failures | | | XXX |
| Pre-fun-in Period | | | xxx |
| Run-in period | | | XXX |
| Randomization failures | | | XXX |
| Randomized | xxx | XXX | XXX |
| Terminated early | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Completed study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Early termination reason | | | |
| Withdrawal by subject | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Investigator / Sponsor Decision | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Randomization Failure | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Lost to follow up | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Non-compliance with Study Procedures | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Screen Failure | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Adverse event | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Protocol deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Pregnancy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Others | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.1.1, 16.2.1.2

N = Total number of randomized subjects in each treatment group. Percentages are based on N.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note:

(1) Percentages for all categories should be based on the number of randomized subjects.

(2) If the column width is not wide enough for the text, do NOT break/truncate the word. Wrap the text around and align with the first text/sentence (i.e. When wrapping, do not allow words to split and indent under the above first letter). This apply to Albabase/Listings.

Table 14.1.2.1 Summary of Protocol Deviations during Pre-run-in Period (All Enrolled Subjects)

| | Number (%) of subjects |
|---|---|
| | Total |
| | (N=xxx) |
| Number of subjects with at least 1 protocol deviation | xxx (xx.x) |
| Total deviations | xxx |
| Exclusion criteria | xxx (xx.x) |
| Inclusion criteria | xxx (xx.x) |
| Informed consent | xxx (xx.x) |

Source: Listing 16.2.2.1

N=Number of subjects screened; percentages are based on N.
The same subject may have had more than 1 protocol deviation.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Notes: Need to verify protocol deviations (from the CRF) occurring during this period - before receiving Run-in treatment

Table 14.1.2.2 Summary of Protocol Deviations during Placebo Run-In Period (Run-in Set)

| | Number (%) of subjects |
|---|---|
| | Total |
| | (N=xxx) |
| Number of subjects with at least 1 protocol deviation | xxx (xx.x) |
| Total deviations | XXX |
| Exclusion criteria | xxx (xx.x) |
| Inclusion criteria | xxx (xx.x) |
| Informed consent | xxx (xx.x) |
| Did not Satisfy Inclusion/Exclusion That May Have<br>Significant Influence on Efficacy (Major PD) [a] | xxx (xx.x) |
| Other deviations | xxx (xx.x) |

Source: Listing 16.2.2.1

Run-in Set: Subjects enrolled in placebo run-in period (between the subjects signing informed consent and administration of the first dose of the randomized study medication) and will be used for presenting run-in period AEs, concomitant medication and protocol deviations.

N=Number of subjects in the run-in population; percentages are based on N.

The same subject may have had more than 1 protocol deviation.

[a] Major PDs occurring in the Run-in period, that contribute to the PP exclusions

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Programming Notes: Need to verify protocol deviations (from the CRF) occurring during this period - run-in period.

Table 14.1.2.3 Summary of Protocol Deviations during Randomized Treatment Period (Safety Analysis Set)

| | Number (%) of subjects | | |
|---|---|---|---|
| | Placebo NS<br>(N=xxx) | GSP 301 NS<br>(N=xxx) | Total<br>(N=xxx) |
| Number of subjects with at least 1 protocol deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Total deviations | XXX | XXX | xxx |
| Concomitant medication | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Exclusion criteria | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Inclusion criteria | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Informed consent | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Study treatment compliance | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Study treatment randomization | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Investigator record keeping source docs | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Study treatment administration/dispense | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Visit scheduling | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not Satisfy Inclusion/Exclusion That May Have Significant Influence on Efficacy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not Treated with Treatment Assigned at Randomization, but Wrongly Treated in Another Treatment Group | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Other Major Deviations | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.2.1

N=Number of subjects in SAS; percentages are based on N.

The same subject may have had more than 1 protocol deviation.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Programming Notes:

<sup>1.</sup> Need to verify protocol deviations (from the CRF) occurring during this period - randomized period.

<sup>2.</sup> If a category above has no data in any of the columns, do not display. New categories might be added at BDRM reviews
Table 14.1.2.4 Summary of Major Protocol Deviations (Safety Analysis Set)

| | | Number (%) of subjects | |
|---|---|---|---|
| | Placebo NS<br>(N=xxx) | GSP 301 NS<br>(N=xxx) | Total<br>(N=xxx) |
| Number of subjects with at least 1 protocol deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| otal deviations | XXX | XXX | XXX |
| Concomitant medication | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Exclusion criteria | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Inclusion criteria | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Informed consent | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Study treatment compliance | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Study treatment randomization | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Investigator record keeping source docs | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Study treatment administration/dispense | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Visit scheduling | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not Satisfy Inclusion/Exclusion That May Have Significant Influence on Efficacy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not Treated with Treatment Assigned at Randomization, but Wrongly Treated in Another Treatment Group | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Other Major Deviations | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.2.1

N=Number of subjects in SAS; percentages are based on N.

The same subject may have had more than 1 major protocol deviation.

## Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Notes:

- 1. Need to verify protocol deviations (all "Major" from the BDRM spreadsheet) regardless of the study period for the SAS subjects.
- 2. If a category above has no data in any of the columns, do not display. New categories might be added at BDRM review.

Table 14.1.3.1 Summary of Analysis Populations

| | | Number (%) of subjects | |
|---|---|---|---|
| | Placebo NS<br>(N=xxx) | GSP 301 NS<br>(N=xxx) | Total<br>(N=xxx) |
| Run-in Set | | | XXX |
| Randomized | xxx | XXX | XXX |
| Not treated as randomized | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not receive any study medication [a] following randomization | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Safety analysis set | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Full analysis set | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Randomized but excluded from FAS | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not receive at least one dose of study medication | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not have at least one post-baseline primary efficacy Assessment | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Randomized twice in the same study [b] | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Per protocol set | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Randomized but excluded from PP due to major protocol deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.1.1, 16.2.3.1, 16.2.3.2

N=Number of subjects randomized; percentages are based on N.

Study medication refers to any study drug taken during the treatment phase of the study [a] Subject who did not receive a study medication is excluded from safety analysis set. [b] <will insert footnote case by case, this line might not be necessary>.

Table 14.1.4.1 Summary of Demographic Data (Run-in Set)

| Demographic characteristic | Statistics | Total |
|---|---|---|
| Characteristic | | (N=xxx) |
| Age (years) | n (%) | xx (xx.x) |
| | Mean (SD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx,xx |
| Age Group (years) n (%) | 6 - < 9 | xxx (xx.x) |
| | 9 - <12 | xxx (xx.x) |
| | Other | xxx (xx.x) |
| | Total | xxx (xx.x) |
| Sex n (%) | Male | xxx (xx.x) |
| | Female | xxx (xx.x) |
| | Total | xxx (xx.x) |
| Race n (%) | White | xxx (xx.x) |
| | African American | xxx (xx.x) |
| | Asian | xxx (xx.x) |
| | American Indian or Alaska Native | xxx (xx.x) |
| | Native Hawaiian or Other Pacific Islander | xxx (xx.x) |
| | Other | xxx (xx.x) |
| | Unknown | xxx (xx.x) |
| | Total | xxx (xx.x) |
| Ethnicity n (%) | Hispanic or Latino | xxx (xx.x) |
| | Not Hispanic or Latino | xxx (xx.x) |
| | Total | xxx (xx.x) |

Run-in Set: Subjects enrolled in placebo run-in period (between the subjects signing informed consent and administration of the first dose of the randomized study medication) and will be used for presenting run-in period AEs, concomitant medication and protocol deviations.

For subject with multiple races, the subject will be counted in each race category.

December 06, 2018

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the treatment Run-in Set group; n= number of subjects with data available; percentages are based on N.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Table 14.1.4.2 Summary of Demographic Data (Safety Analysis Set)

| Demographic | Statistics | Placebo NS | GSP 301 NS | Total |
|---|---|---|---|---|
| characteristic | Statistics | (N=xxx) | (N=xxx) | (N=xxx) |
| Age (years) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | XX.X |
| | Min, Max | xx,xx | xx,xx | xx,xx |
| Age Group (years) n (%) | 6 - < 9 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | 9 - <12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Other | xxx (xx.x) | , , | (, |
| | Total | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Sex n (%) | Male | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Female | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Race n (%) | White | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | African American | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Asian | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | American Indian or Alaska Native | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Native Hawaiian or Other Pacific Islander | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Other | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Unknown | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Ethnicity n (%) | Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Not Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Total | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

For subject with multiple races, the subject will be counted in each race category.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in SAS in the treatment group; n= number of subjects with data available; percentages are based on N.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Table 14.1.4.3 Summary of Demographic Data (Full Analysis Set) Repeat table 14.1.4.1 for Full Analysis Set

Table 14.1.4.4 Summary of Demographic Data (Per Protocol Set) Repeat table 14.1.4.1 for Per Protocol Set.

Table 14.2.1.1 Summary of Average AM and PM rTNSS by Day (Full Analysis Set)

| | | | Average AM an | d PM rTNSS | by Day | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Day | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| Placebo NS ( $N = xxx$ ) | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | XX | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |
| GSP 301 NS $(N = xxx)$ | Baseline | XX | xx.x (xx. x) | XX.X | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments, and so on for the rest of the treatment.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Table 14.2.1.2 Summary of Repeated Measures Analysis Results of Average AM and PM rTNSS over the 14-day Treatment Period (Full Analysis Set)

Overall 14-day treatment period

| | | n | LS M | LS Mean (SE) | | Comparison between GSP 301 NS vs. Placebo NS | | |
|---|---|---|---|---|---|---|---|---|
| Treatment Group Comparison (GSP 301 NS vs. Placebo NS) | Placebo<br>NS | GSP 301<br>NS | Placebo<br>NS | GSP 301<br>NS | LS Mean<br>Difference | SE of LS Mean<br>Difference | 95% CI | P-value |
| GSP 301 NS vs. Placebo NS | xxx | XXX | xxx.x<br>(xx.xx) | xxx.x<br>(xx.xx) | xxx.x | xxx.xx | (xxx.x, xxx.x) | X.XXX |

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Notes:

- 1. Repeat the analysis for Days 1 to 14, replacing "Overall 14-day treatment period" with "Day 1", "Day 2", as is appropriate
- 2. Based on the results of the independent modeling for interactions, add the following footnotes:
  - a. If only treatment\*site interaction is significant, footnote: "Site by treatment interaction is included in the model for the Overall 14-day analysis".
  - b. If only baseline\*treatment interaction is significant, footnote: "Baseline score by treatment interaction is included in the model for the Overall 14-day analysis".
  - c. If both interactions are significant, footnote: "Site by treatment and baseline score by treatment interactions are included in the model for the Overall I4-day analysis".

Table 14.2.1.3 Summary of Average AM and PM rTNSS by Day (Per Protocol Set)

Source: Listing 16.2.6.3

Repeat Table 14.2.1.1 for per protocol set.

Table 14.2.1.4 Summary of Repeated Measures Analysis Results of Average AM and PM rTNSS over the 14-day Treatment Period (Per Protocol Set)

Source: Listing 16.2.6.3

Repeat Table 14.2.1.2 for per protocol set.

Table 14.2.1.5 Subgroup Analyses (Age Group): Summary of Average AM and PM rTNSS by Day (Full Analysis Set)

Age Group 6 - <9

| | | | Average AM and | d PM rTNSS | by Day | | Change | from Baselin | ne |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Day | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| Placebo NS (N = xxx) | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | XX | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |
| GSP 301 NS $(N = xxx)$ | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x(xx.x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX,X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | XX | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Repeat for Age Group 9-<12.

Table 14.2.1.6 Subgroup Analyses (Age Group): Summary of Repeated Measures Analysis Results of Average AM and PM rTNSS over the 14-day Treatment Period (Full Analysis Set)

Age Group: 6-<9

Overall 14-day treatment period

| | | n | LS Mean (SE) | | Comparison between GSP 301 NS vs. Placebo NS | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment Group Comparison | Placebo | GSP 301 | Placebo | GSP 301 | LS Mean | SE of LS Mean | | |
| (GSP 301 NS vs. Placebo NS) | NS | NS | NS | NS | Difference | Difference | 95% CI | P-value |
| GSP 301 NS vs. Placebo NS | xxx | xxx | xxx.x<br>(xx.xx) | xxx.x<br>(xx.xx) | XXX.X | xxx.xx | (xxx.x, xxx.x) | x.xxx |

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Notes:

- 1. Repeat the analysis for Days 1 to 14, replacing "Overall 14-day treatment period" with "Day 1", "Day 2", as is appropriate
- 2. Based on the results of the independent modeling for interactions, add the following footnotes:
  - a. If only treatment\*site interaction is significant, footnote: "Site by treatment interaction is included in the model for the Overall 14-day analysis".
  - b. If only baseline\*treatment interaction is significant, footnote: "Baseline score by treatment interaction is included in the model for the Overall 14-day analysis".
  - c. If both interactions are significant, footnote: "Site by treatment and baseline score by treatment interactions are included in the model for the Overall 14-day analysis".
- 3. Repeat the analysis for Age Group 9-<12.

Table 14.2.1.7 Subgroup Analyses (Sex): Summary of Average AM and PM rTNSS by Day (Full Analysis Set)

Sex: Male

| | | | Average AM and | d PM rTNSS | by Day | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Day | n | Mean (SD) | Median | Min, Max | п | Mean (SD) | Median | Min, Max |
| Placebo NS (N = xxx) | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | XX | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |
| GSP 301 NS $(N = xxx)$ | Baseline | XX | xx.x (xx. x) | XX.X | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | xx | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Repeat for Sex: Female.

Table 14.2.1.8 Subgroup Analyses (Race): Summary of Average AM and PM rTNSS by Day (Full Analysis Set)

Race: White

| | | | Average AM and | d PM rTNSS | by Day | | Change | from Baselii | ne |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Day | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| Placebo NS ( $N = xxx$ ) | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| GSP 301 NS $(N = xxx)$ | Baseline | xx | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | XX | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

For subject with multiple races, the subject will be included in each race subgroup analysis.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYYY HH:MM

Repeat for each race: White, African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Other.

Table 14.2.1.9 Subgroup Analyses (Ethnicity): Summary of Average AM and PM rTNSS by Day (Full Analysis Set)

Ethnicity: Hispanic or Latino

| | | | Average AM and | d PM rTNSS | by Day | | Change: | from Baselin | ne |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Day | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| Placebo NS (N = xxx) | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x(xx.x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | xx | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |
| GSP 301 NS (N = xxx) | Baseline | xx | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x(xx.x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | xx | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Repeat for Not Hispanic or Latino

Table 14.2.2.1.1 Summary of Average AM and PM iTNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.4

Repeat table 14.2.1.1 for iTNSS, replace spanner label < rTNSS by Day> with <iTNSS by Day>

Table 14.2.2.1.2 Summary of Repeated Measures Analysis Results of Average AM and PM iTNSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.4

Repeat table 14.2.1.2 for iTNSS

Table 14.2.2.1.3 Summary of Average AM and PM iTNSS by Day (Per Protocol Set)

Source: Listing 16.2.6.4

Repeat table 14.2.1.3 for iTNSS, replace spanner label < rTNSS by Day> with <iTNSS by Day>

Table 14.2.2.1.4 Summary of Repeated Measures Analysis Results of Average AM and PM iTNSS over the 14-day Treatment Period (Per Protocol Set)

Source: Listing 16.2.6.4

Repeat table 14.2.1.4 for iTNSS

Table 14.2.2.1.5 Subgroup Analyses (Age Group): Summary of Average AM and PM iTNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.4

 $\textit{Repeat table 14.2.1.5 for iTNSS, replace spanner label} < \textit{rTNSS by Day} > \textit{with} < \textit{iTNSS by Day} > \textit{one of the property of the prope$ 

Table 14.2.2.2.1 Summary of Average AM and PM rTOSS by Day (Full Analysis Set)

Source: Listing 16.2.6.9

Repeat table 14.2.1.1 for rTOSS, replace spanner label < rTNSS by Day> with <rTOSS by Day>

Table 14.2.2.2.2 Summary of Repeated Measures Analysis Results of Average AM and PM rTOSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.9

Repeat table 14.2.1.2 for rTOSS

Table 14.2.2.2.3 Summary of Average AM and PM rTOSS by Day (Per Protocol Set)

Source: Listing 16.2.6.9

Repeat table 14.2.1.3 for rTOSS, replace spanner label < rTNSS by Day> with <rTOSS by Day>

Table 14.2.2.2.4 Summary of Repeated Measures Analysis Results of Average AM and PM rTOSS over the 14-day Treatment Period (Per Protocol Set)

Source: Listing 16.2.6.9

Repeat table 14.2.1.4 for rTOSS

Table 14.2.2.2.5 Subgroup Analyses (Age Group): Summary of Average AM and PM rTOSS by Day (Full Analysis Set)

Source: Listing 16.2.6.9

Repeat table 14.2.1.5 for rTOSS, replace spanner label < rTNSS by Day> with <rTOSS by Day>

Table 14.2.2.3.1 Summary of the Overall PRQLQ Score and Individual Domains on Day 15 (Full Analysis Set)

| PRQLQ Domain | | Statistics | Placebo NS | GSP 301 NS | Total |
|---|---|---|---|---|---|
| FRQLQ Dollialli | | Statistics | (N=xxx) | (N=xxx) | (N=xxx) |
| Overall PRQLQ | Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | xx.x | XX.X |
| | | Min, Max | xx,xx | xx,xx | xx,xx |
| | Day 15 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | xx.x |
| | | Min, Max | xx,xx | xx,xx | xx,xx |
| | Change from Baseline to Day 15 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | - | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | xx.x |
| | | Min, Max | xx,xx | xx,xx | xx,xx |
| PRQLQ Domain<br>Activity Limitations<br>Practical Problems | | | | | |
| Nose Symptoms | | | | | |
| Eye Symptoms | | | | | |
| Other Symptoms | | | | | |

Source: Listing 16.2.6.11

Baseline is defined as the time point "pre-dosing" at the Randomization Visit (Visit 2). Day 15 includes Visit 4 for all subjects, including those terminating early, regardless of what actual study day this visit occurred on.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat the summary for each domain as listed in the table

Table 14.2.2.3.2 Summary of ANCOVA Analysis Results of the Overall PRQLQ Score and Individual Domains on Day 15 (Full Analysis Set)

Overall PRQLQ

| | 1 | n | LS M | ean (SE) | Compari | son between GSP | 301 NS and Place | bo NS |
|---|---|---|---|---|---|---|---|---|
| Treatment Group Comparison (GSP 301 NS vs. Placebo NS) | Placebo<br>NS | GSP 301<br>NS | Placebo<br>NS | GSP 301<br>NS | LS Mean<br>Difference | SE of LS Mean<br>Difference | 95% CI | P-value |
| GSP 301 NS vs. Placebo NS | XXX | XXX | xxx.x<br>(xx.xx) | xxx.x<br>(xx.xx) | xxx.x | xxx.xx | (xxx.x, xxx.x) | X.XXX |

Source: Listing 16.2.6.11

Baseline is defined as the time point "pre-dosing" at the Randomization Visit (Visit 2). Day 15 includes Visit 4 for all subjects, including those terminating early, regardless of what actual study day this visit occurred on.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: analysis of covariance (ANCOVA) with change from baseline as dependent variable, treatment group and site as fixed effect and baseline as covariate.

Individual statistical analysis models were made separately for each of the PRQLQ domains.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

## Programming Note:

- 1. Repeat the analysis for each domain listed in table 14.2.2.3.1, replacing "Overall PRQLQ" with the domain name as is appropriate
- 2. Based on the results of the independent modeling for interactions, add the following footnotes:
  - a. If only treatment\*site interaction is significant, footnote: "Site by treatment interaction is included in the model for the Overall PRQLQ analysis".
  - b. If only baseline\*treatment interaction is significant, footnote: "Baseline score by treatment interaction is included in the model for the Overall PRQLQ analysis".
  - c. If both interactions are significant, footnote: "Site by treatment and baseline score by treatment interactions are included in the model for the Overall PRQLQ analysis".

Table 14.2.2.3.3 Subgroup Analysis (Age Group): Summary of the Overall PRQLQ Score and Individual Domains on Day 15 (Full Analysis Set)

Age Group: 6-<9

| PRQLQ Domain | | Statistics | Placebo NS<br>(N=xxx) | GSP 301 NS<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|
| Overall PRQLQ | Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | XX.X |
| | | Min, Max | xx,xx | xx,xx | xx,xx |
| | Day 15 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | XX.X |
| | | Min, Max | xx,xx | xx,xx | xx,xx |
| | Change from Baseline to Day 15 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | • | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | xx.x |
| | | Min, Max | XX,XX | xx,xx | XX,XX |

Baseline is defined as the time point "pre-dosing" at the Randomization Visit (Visit 2). Day 15 includes Visit 4 for all subjects, including those terminating early, regardless of what actual study day this visit occurred on.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat the summary for age group 9-<12.

Table 14.2.3.1.1 Summary of AM rTNSS by Day (Full Analysis Set)

| | | | Average AN | 1 rTNSS by I | Day | | Change: | from Baselin | ne |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Day | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| Placebo NS (N = xxx) | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 2 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x(xx.x) | XX.X | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 15 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| GSP 301 NS $(N = xxx)$ | Baseline | XX | xx.x (xx. x) | XX.X | (xx,xx) | | | | |
| | 2 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 15 | xx | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |

Baseline score is derived as the mean of the last 4 consecutive AM values prior to randomization, during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Table 14.2.3.1.2 Summary of Repeated Measures Analysis Results of AM rTNSS over the 14-day Treatment Period (Full Analysis Set)

| Overall 14-day treatr | nent period |
|-----------------------|-------------|
|-----------------------|-------------|

| | | n | LS M | lean (SE) | Compari | son between GSP: | 301 NS and Place | bo NS |
|---|---|---|---|---|---|---|---|---|
| Treatment Group Comparison (GSP 301 NS vs. Placebo NS) | Placebo<br>NS | GSP 301<br>NS | Placebo<br>NS | GSP 301<br>NS | LS Mean<br>Difference | SE of LS Mean<br>Difference | 95% CI | P-value |
| GSP 301 NS vs. Placebo NS | XXX | XXX | xxx.x<br>(xx.xx) | xxx.x<br>(xx.xx) | XXX.X | xxx.xx | (xxx.x, xxx.x) | x.xxx |

Baseline score is derived as the mean of the last 4 consecutive AM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Day is an unordered categorical variable and Treatment by Day interaction is fitted in the model for the Day 2 to Day 15 analyses.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Notes: Repeat the analysis for Days 2 to 15, replacing "Overall 14-day treatment period" with "Day 2", "Day 3", as is appropriate

Table 14.2.3.2.1 Summary of PM rTNSS by Day (Full Analysis Set)

Repeat table 14.2.3.1.1 for PM rTNSS; replace spanner label <Average AM rTNSS by Day> with <Average PM rTNSS by Day>, Days will go from 1 to 14.

Change footnote to:

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 4 consecutive PM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available

Table 14.2.3.2.2 Summary of Repeated Measures Analysis Results of PM rTNSS over the 14-day Treatment Period (Full Analysis Set)

Repeat table 14.2.3.1.2 for PM rTNSS

Change footnote to:

Source: Listing 16.2.6.3

Baseline score is derived as the mean of the last 4 consecutive PM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Day is an unordered categorical variable and Treatment by Day interaction is fitted in the model for the Day 1 to Day 14 analyses.

Programming Notes: Repeat the analysis for Days 1 to 14, replacing "Overall 14-day treatment period" with "Day 1", "Day 2", as is appropriate

Table 14.2.3.3.1 Summary of AM iTNSS by Day (Full Analysis Set)

Repeat table 14.2.3.1.1 for iTNSS, replace spanner label < rTNSS by Day> with <iTNSS by Day>

Change footnote to:

Source: Listing 16.2.6.4

Baseline score is derived as the mean of the last 4 consecutive AM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Table 14.2.3.3.2 Summary of Repeated Measures Analysis Results of AM iTNSS over the 14-day Treatment Period (Full Analysis Set)

Repeat table 14.2.3.1.2 for iTNSS, replace spanner label < rTNSS by Day> with <iTNSS by Day>

Change footnote to: Source: Listing 16.2.6.4

Baseline score is derived as the mean of the last 4 consecutive AM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Day is an unordered categorical variable and Treatment by Day interaction is fitted in the model for the Day 2 to Day 15 analyses.

Table 14.2.3.4.1 Summary of PM iTNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.4

Repeat table 14.2.3.2.1 for iTNSS, replace spanner label < rTNSS by Day> with <iTNSS by Day>

Change footnote to:

Baseline score is derived as the mean of the last 4 consecutive PM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Table 14.2.3.4.2 Summary of Repeated Measures Analysis Results of PM iTNSS over the 14-day Treatment Period (Full Analysis Set)

Change footnote to:

Source: Listing 16.2.6.4

Baseline score is derived as the mean of the last 4 consecutive PM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Day is an unordered categorical variable and Treatment by Day interaction is fitted in the model for the Day 1 to Day 14 analyses.

Table 14.2.3.5.1 Summary of Average AM and PM Reflective Individual Nasal Symptoms by Day (Full Analysis Set)

Symptom: Nasal Congestion

| | | | Average AM ar | d PM score l | by Day | | Change | from Baselir | ne |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Day | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| Placebo NS (N = xxx) | Baseline | XX | xx.x (xx. x) | xx.x | (xx,xx) | | | | |
| | 1 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x(xx.x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | xx.x | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | xx.x | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | xx | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | XX.X | (xx,xx) |
| GSP 301 NS $(N = xxx)$ | Baseline | XX | xx.x (xx. x) | XX.X | (xx,xx) | | | | |
| | 1 | XX | xx.x(xx.x) | XX.X | (xx,xx) | XX | xx.x(xx.x) | XX.X | (xx,xx) |
| | 2 | XX | xx.x(xx.x) | XX.X | (xx,xx) | XX | xx.x(xx.x) | xx.x | (xx,xx) |
| | 3 | XX | xx.x (xx. x) | XX.X | (xx,xx) | XX | xx.x (xx. x) | XX.X | (xx,xx) |
| | 14 | xx | xx.x (xx. x) | xx.x | (xx,xx) | xx | xx.x (xx. x) | xx.x | (xx,xx) |

Source: Listing 16.2.6.1

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat table for each symptom; Nasal congestion, Rhinorrhea, Nasal Itching, Sneezing

Table 14.2.3.5.2 Summary of Repeated Measures Analysis Results of Average AM and PM Reflective Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set)

Symptom: Nasal Congestion

| | | n | LS Mean (SE) Comparison between GSP 301 | | 301 NS and Place | 1 NS and Placebo NS | | |
|---|---|---|---|---|---|---|---|---|
| Treatment Group Comparison (GSP 301 NS vs. Placebo NS) | Placebo<br>NS | GSP 301<br>NS | Placebo<br>NS | GSP 301<br>NS | LS Mean<br>Difference | SE of LS Mean<br>Difference | 95% CI | P-value |
| GSP 301 NS vs. Placebo NS | xxx | xxx | xxx.x<br>(xx.xx) | xxx.x<br>(xx.xx) | XXX.X | xxx.xx | (xxx.x, xxx.x) | X.XXX |

Source: Listing 16.2.6.1

Baseline score is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization. Day 1 is derived as the average of Day 1 PM and Day 2 AM assessments and so on for the rest of the treatment period.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Notes: Overall 14-day treatment period only, repeat table for each symptom; Nasal congestion, Rhinorrhea, Nasal Itching, Sneezing

Table 14.2.3.6.1 Summary of AM Reflective Individual Nasal Symptoms by Day (Full Analysis Set)

Repeat table 14.2.3.5.1 for AM rTNSS; replace spanner label < Average AM and PM score by Day> with <AM score by Day>

Change footnote to:

Source: Listing 16.2.6.1

Baseline score is derived as the mean of the last 4 consecutive AM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available

Table 14.2.3.6.2 Summary of Repeated Measures Analysis Results of AM Reflective Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set)

Repeat table 14.2.3.5.2 for AM rTNSS

Change footnote to:

Source: Listing 16.2.6.1

Baseline score is derived as the mean of the last 4 consecutive AM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Table 14.2.3.7.1 Summary of PM Reflective Individual Nasal Symptoms by Day (Full Analysis Set)

Repeat table 14.2.3.5.1 for PM rTNSS; replace spanner label < Average AM and PM score by Day> with <PM score by Day>

Change footnote to:

Source: Listing 16.2.6.1

Baseline score is derived as the mean of the last 4 consecutive PM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available

Table 14.2.3.7.2 Summary of Repeated Measures Analysis Results of PM Reflective Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set)

Repeat table 14.2.3.5.2 for PM rTNSS

Change footnote to:

Source: Listing 16.2.6.1

Baseline score is derived as the mean of the last 4 consecutive PM values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: Mixed-effect repeated measures model with change from baseline as the dependent variable, treatment group and site as fixed effects, baseline score as covariate and study day as the within-subject effect.

Table 14.2.3.8.1 Summary of Average AM and PM Instantaneous Individual Nasal Symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.2

Repeat table 14.2.3.5.1 for Instantaneous Individual Nasal Symptoms including itching/burning eyes, tearing/watering eyes

Table 14.2.3.8.2 Summary of Repeated Measures Analysis Results of Average AM and PM Instantaneous Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.2

Repeat table 14.2.3.5.2 for Instantaneous Individual Nasal Symptoms

Table 14.2.3.9.1 Summary of AM Instantaneous Individual Nasal Symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.2

Repeat table 14.2.3.6.1 for Instantaneous Individual Nasal Symptoms

Table 14.2.3.9.2 Summary of Repeated Measures Analysis Results of AM Instantaneous Individual Nasal Symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.2

Repeat table 14.2.3.6.2 for Instantaneous Individual Nasal Symptoms

Table 14.2.3.10.1 Summary of PM Instantaneous Individual Nasal Symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.2

Repeat table 14.2.3.7.1 for Instantaneous Individual Nasal Symptoms

Table 14.2.3.10.2 Summary of Repeated Measures Analysis Results of PM Instantaneous Individual Nasal Symptoms over the 14-day Treatment Period (Full

Analysis Set)

Source: Listing 16.2.6.2

Repeat table 14.2.3.57.2 for Instantaneous Individual Nasal Symptoms

Table 14.2.3.11.1 Summary of Average AM and PM iTOSS by Day (Full Analysis Set)

Source: Listing 16.2.6.10

Repeat table 14.2.2.1.1 for iTOSS, replace spanner label < iTNSS by Day> with <iTOSS by Day>

Table 14.2.3.11.2 Summary of Repeated Measures Analysis Results of Average AM and PM iTOSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.10

Repeat table 14.2.2.1.2 for iTOSS

Table 14.2.3.12.1 Summary of AM rTOSS by Day (Full Analysis Set)

Source: Listing 16.2.6.9

Repeat table 14.2.3.1.1 for AM rTOSS; replace spanner label <rTNSS by Day> with <rTOSS by Day>

Table 14.2.3.12.2 Summary of Repeated Measures Analysis Results of AM rTOSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.9

Repeat table 14.2.3.1.2 for AM rTOSS

Table 14.2.3.13 1 Summary of PM rTOSS by Day (Full Analysis Set)

Source: Listing 16.2.6.9

Repeat table 14.2.3.1.1 for PM rTOSS; replace spanner label <Average AM rTNSS by Day> with < Average PM rTOSS by Day>

Table 14.2.3.13 2 Summary of Repeated Measures Analysis Results of PM rTOSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.9

Repeat table 14.2.3.1.2 for PM rTOSS

Table 14.2.3.14.1 Summary of AM iTOSS by Day (Full Analysis Set)

Source: Listing 16.2.6.10

Repeat table 14.2.3.1.1 for AM iTOSS; replace spanner label <rTNSS by Day> with <iTOSS by Day>

Table 14.2.3.14.2 Summary of Repeated Measures Analysis Results of AM iTOSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.10

Repeat table 14.2.3.1.2 for AM iTOSS

Table 14.2.3.15.1 Summary of PM iTOSS by Day (Full Analysis Set)

Source: Listing 16.2.6.10

Repeat table 14.2.3.1.1 for PM iTOSS; replace spanner label <Average AM rTNSS by Day> with <Average PM iTOSS by Day>

Table 14.2.3.15.2 Summary of Repeated Measures Analysis Results of PM iTOSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.10

Repeat table 14.2.3.1.2 for PM iTOSS

Table 14.2.3.16.1 Summary of Average AM and PM rTNNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.7

Repeat table 14.2.2.1.1 for rTNNSS, replace spanner label < iTNSS by Day> with <rTNNSS by Day>

Table 14.2.3.16.2 Summary of Repeated Measures Analysis Results of Average AM and PM rTNNSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.7

Repeat table 14.2.2.1.2 for rTNNSS

Table 14.2.3.17.1 Summary of Average AM and PM iTNNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.8

Repeat table 14.2.2.1.1 for iTNNSS, replace spanner label < iTNSS by Day > with <iTNNSS by Day >

Table 14.2.3.17.2 Summary of Repeated Measures Analysis Results of Average AM and PM iTNNSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.8

Repeat table 14.2.2.1.2 for iTNNSS

Table 14.2.3.18.1 Summary of AM rTNNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.7

Repeat table 14.2.3.1.1 for AM rTNNSS; replace spanner label <rTNSS by Day> with <rTNNSS by Day>

Table 14.2.3.18.2 Summary of Repeated Measures Analysis Results of AM rTNNSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.7

Repeat table 14.2.3.1.2 for AM rTNNSS

Table 14.2.3.19.1 Summary of PM rTNNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.7

Repeat table 14.2.3.1.1 for PM rTNNSS; replace spanner label <Average AM rTNSS by Day> with < Average PM rTNNSS by Day>

Table 14.2.3.19.2 Summary of Repeated Measures Analysis Results of PM rTNNSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.7

Repeat table 14.2.3.1.2 for PM rTNNSS

Table 14.2.3.20.1 Summary of AM iTNNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.8

Repeat table 14.2.3.1.1 for AM iTNNSS; replace spanner label <rTNSS by Day> with <iTNNSS by Day>

Table 14.2.3.20.2 Summary of Repeated Measures Analysis Results of AM iTNNSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.8

Repeat table 14.2.3.1.2 for AM iTNNSS

Table 14.2.3.21.1 Summary of PM iTNNSS by Day (Full Analysis Set)

Source: Listing 16.2.6.8

Repeat table 14.2.3.1.1 for PM iTNNSS; replace spanner label <Average AM rTNSS by Day> with < Average PM iTNNSS by Day>

Table 14.2.3.21.2 Summary of Repeated Measures Analysis Results of PM iTNNSS over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.8

Repeat table 14.2.3.1.2 for PM iTNNSS

Table 14.2.3.22.1 Summary of Average AM and PM Reflective Individual Non-nasal symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.5

Repeat table 14.2.3.5.1 for Reflective Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.22.2 Summary of Repeated Measures Analysis Results of Average AM and PM Reflective Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.5

Repeat table 14.2.3.5.2 for Reflective Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.23.1 Summary of AM Reflective Individual Non-nasal symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.5

Repeat table 14.2.3.6.1 for Reflective Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.23.2 Summary of Repeated Measures Analysis Results of AM Reflective Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.5

Repeat table 14.2.3.6.2 for Reflective Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.24.1 Summary of PM Reflective Individual Non-nasal symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.5

Repeat table 14.2.3.7.1 for Reflective Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.24.2 Summary of Repeated Measures Analysis Results of PM Reflective Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.5

Repeat table 14.2.3.7.2 for Reflective Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.25.1 Summary of Average AM and PM instantaneous Individual Non-nasal symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.6

Repeat table 14.2.3.5.1 for instantaneous Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.25.2 Summary of Repeated Measures Analysis Results of Average AM and PM instantaneous Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.6

Repeat table 14.2.3.5.2 for instantaneous Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of
Ears or Palate

Table 14.2.3.26.1 Summary of AM instantaneous Individual Non-nasal symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.6

Repeat table 14.2.3.6.1 for instantaneous Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of
Ears or Palate

Table 14.2.3.26.2 Summary of Repeated Measures Analysis Results of AM instantaneous Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.6

Repeat table 14.2.3.6.2 for instantaneous Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of
Ears or Palate

Table 14.2.3.27.1 Summary of PM instantaneous Individual Non-nasal symptoms by Day (Full Analysis Set)

Source: Listing 16.2.6.6

Repeat table 14.2.3.7.1 for instantaneous Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.27.2 Summary of Repeated Measures Analysis Results of PM instantaneous Individual Non-nasal symptoms over the 14-day Treatment Period (Full Analysis Set)

Source: Listing 16.2.6.6

Repeat table 14.2.3.7.2 for instantaneous Individual Non-nasal symptoms including itching/burning eyes, tearing/watering eyes, redness of eyes and Itching of Ears or Palate

Table 14.2.3.28.1 Summary of Physician Assessed Nasal Symptoms Score (PNSS) and Individual Assessments at Day 15 (Full Analysis Set)

| | | | Placebo NS | GSP 301 NS | Total |
|---|---|---|---|---|---|
| Symptom | | Statistics | (N=xxx) | (N=xxx) | (N=xxx) |
| Overall PNSS Score | Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx,xx | xx,xx | xx,xx |
| | Day 15 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | xx.x | xx.x |
| | | Min, Max | xx,xx | xx,xx | xx,xx |
| | Change from Baseline to Day 15 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | - | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X | xx.x |
| | | Min, Max | xx,xx | xx,xx | xx,xx |

Individual Symptoms: Rhinorrhea Nasal Congestion Nasal Itching Sneezing

Source: Listing 16.2.6.12

Baseline is defined as the time point "pre-dosing" at the Randomization Visit (Visit 2).

Day 15 includes Visit 4 for all subjects, including those terminating early, regardless of what actual study day this visit occurred on.

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the FAS treatment group; n= number of subjects with data available

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat the summary for each symptom as listed in the table

Table 14.2.3.28.2 Summary of ANCOVA Analysis Results of Physician Assessment of Nasal Symptoms Score (PNSS) and individual assessments at Day 15 (Full Analysis Set)

## Overall PNSS

| | | n | LS Mean (SE) | | Comparison between GSP 301 NS and Placebo NS | | | bo NS |
|---|---|---|---|---|---|---|---|---|
| Treatment Group Comparison | Placebo | GSP 301 | Placebo | GSP 301 | LS Mean | SE of LS Mean | | |
| (GSP 301 NS vs. Placebo NS) | NS | NS | NS | NS | Difference | Difference | 95% CI | P-value |
| GSP 301 NS vs. Placebo NS | xxx | xxx | xxx.x<br>(xx.xx) | xxx.x<br>(xx.xx) | XXX.X | xxx.xx | (xxx.x, xxx.x) | X.XXX |

Source: Listing 16.2.6.12

Baseline is defined as the time point "pre-dosing" at the Randomization Visit (Visit 2). Day 15 includes Visit 4 for all subjects, including those terminating early, regardless of what actual study day this visit occurred on.

n= number of subjects with data available LS = least squares; SE = standard error

Statistical Analysis model: analysis of covariance (ANCOVA) with change from baseline as dependent variable, treatment group and site as fixed effect and baseline as covariate.

Individual statistical analysis models were made separately for each of the PNSS individual symptoms.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat the analysis for each symptom listed in table 14.2.3.28.1, replacing "Overall PNSS" with the symptom as is appropriate

Table 14.3.1.1 Overall Summary of Treatment Emergent Adverse Event (TEAE) (Safety Analysis Set)

| | Placebo NS | GSP 301 NS |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| | n (%) | n (%) |
| Number of subjects with any treatment-emergent adverse event[a] | xxx (xx.x) | xxx (xx.x) |
| Any related treatment-emergent adverse event | , | |
| Any treatment-emergent severe adverse event | xxx (xx.x) | xxx (xx.x) |
| Any treatment-emergent moderate adverse event | xxx (xx.x) | xxx (xx.x) |
| Any treatment-emergent mild adverse event | xxx (xx.x) | xxx (xx.x) |
| Any treatment-emergent SAE leading to death | xxx (xx.x) | xxx (xx.x) |
| Any treatment-emergent SAE (including events leading to death) | xxx (xx.x) | xxx (xx.x) |
| Any treatment-emergent adverse event leading to study | xxx (xx.x) | xxx (xx.x) |
| discontinuation | | |
| Number of treatment-emergent adverse events [b] | XXX | xxx |
| Severity | | |
| Mild | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) |
| Severe | xxx (xx.x) | xxx (xx.x) |
| Relationship | | |
| Related | xxx (xx.x) | xxx (xx.x) |
| Not Related | xxx (xx.x) | xxx (xx.x) |
| TEAE leading to study discontinuation | xxx (xx.x) | xxx (xx.x) |
| TEAEs leading to death | xxx (xx.x) | xxx (xx.x) |
| Treatment-emergent SAEs (including events leading to death) | xxx (xx.x) | xxx (xx.x) |
| Related treatment-emergent SAEs | xxx (xx.x) | xxx (xx.x) |

Program: xxxx.sas Executed: DDMMMYYYYY HH:MM

<sup>[</sup>a] Subjects with multiple events in the same category are counted only once in that category. Subjects with events in more than 1 category are counted once in each of those categories. Percentages are based on total number of subjects in the safety set within each treatment group.

<sup>[</sup>b] Percentages in the succeeding categories are based on the number of treatment-emergent adverse events.
Table 14.3.1.2 Summary of Treatment-Emergent Adverse Events (Safety Analysis Set)

| System Organ Class | Placebo (N=xxx | | GSP 301 NS<br>(N=xxx) | |
|---|---|---|---|---|
| Preferred Term | Number (%) of subjects[a] | Event Rate[b] | Number (%) of subjects[a] | Event Rate[b] |
| Number of treatment-emergent adverse events | xxx | | xxx | |
| Number of subjects with any treatment-emergent adverse event | xxx (xx.x) | x.xx | xxx (xx.x) | x.xx |
| System Organ Class # 1 | xxx (xx.x) | x.xx | xxx (xx.x) | x.xx |
| Preferred Term # 1 | xxx (xx.x) | x.xx | xxx (xx.x) | x.xx |
| Preferred Term # 2 | xxx (xx.x) | x.xx | xxx (xx.x) | x.xx |
| 89%. | | | | |
| System Organ Class # 2 | xxx (xx.x) | x.xx | xxx (xx.x) | x.xx |
| Preferred Term # 1 | xxx (xx.x) | x.xx | xxx (xx.x) | X.XX |
| Preferred Term # 2 | xxx (xx.x) | X.XX | xxx (xx.x) | x.xx |
| 600 | | | | |

Source: Listing 16.2.7.1

N= Number of subjects in SAS treatment arm; percentages are based on N.

[a] Number (%) of subjects with AEs, sorted on international order for system organ class and alphabetically for preferred term.

[b] Number of subjects with AEs divided by the total duration (day) of treatment across all subjects in given treatment group, multiplied by 100.

The total number of TEAEs counts all treatment-emergent AEs for subjects. At each level of subject summarization, a subject is counted once if the subject reported one or more events.

Adverse Events were coded using MedDRA, Version 21.0.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: For event rate, the denominator is total duration in days of treatment for all subjects in the treatment group.

109

Table 14.3.1.3 Summary of Treatment-Related Emergent Adverse Events (Safety Analysis Set)

Source: Listing 16.2.7.1

Repeat table 14.3.1.2 for treatment-related adverse events

Table 14.3.1.4 Summary of Treatment-Emergent Adverse Events Leading to Discontinuation (Safety Analysis Set)

Source: Listing 16.2.7.4

Repeat table 14.3.1.2 for TEAEs leading to discontinuation

Table 14.3.1.5 Summary of Treatment-Emergent Adverse Events by Severity (Safety Analysis Set)

| System Organ Class | Placebo NS | GSP 301 NS |
|---|---|---|
| Preferred Term | (N=xxx) | (N=xxx) |
| Severity | n (%) | n (%) |
| Number of treatment-emergent adverse events | XXX | xxx |
| Mild | xxx | XXX |
| Moderate | XXX | XXX |
| Severe | xxx | xxx |
| Number of subjects with any treatment-emergent adverse event | xxx (xx.x) | xxx (xx.x) |
| Mild | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) |
| Severe | xxx (xx.x) | xxx (xx.x) |
| System Organ Class # 1 | xxx (xx.x) | xxx (xx.x) |
| Mild | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) |
| severe | xxx (xx.x) | xxx (xx.x) |
| Preferred Term # 1 | xxx (xx.x) | xxx (xx.x) |
| Mild | xxx (xx.x) | xxx (xx.x) |
| 3699 | | |

Source: Listing 16.2.7.1

N= Number of subjects in SAS treatment arm, percentages are based on N.

The total number of TEAEs counts all treatment-emergent AEs for subjects. At each level of subject summarization, a subject is counted once for the most severe event if the subject reported one or more events.

If the severity of an adverse event is missing, the AE is reported as "Severe".

Adverse Events were coded using MedDRA, Version 21.0.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Table 14.3.1. 6 Summary of Treatment-Emergent Adverse Events by Relationship to Study Treatment (Safety Analysis Set)

| System Organ Class | Placebo NS | GSP 301 NS |
|---|---|---|
| Preferred Term | (N=xxx) | (N=xxx) |
| Relationship | n (%) | n (%) |
| Number of treatment-emergent adverse events | xxx | xxx |
| Not Related | XXX | XXX |
| Related | xxx | xxx |
| Number of subjects with any treatment-emergent adverse event | xxx (xx.x) | xxx (xx.x) |
| Not Related | xxx (xx.x) | xxx (xx.x) |
| Related | xxx (xx.x) | xxx (xx.x) |
| System Organ Class # 1 | xxx (xx.x) | xxx (xx.x) |
| Not Related | xxx (xx.x) | xxx (xx.x) |
| Related | xxx (xx.x) | xxx (xx.x) |
| Preferred Term # 1 | xxx (xx.x) | xxx (xx.x) |
| Not Related | xxx (xx.x) | xxx (xx.x) |
| Related | xxx (xx.x) | xxx (xx.x) |
| | , | |

Source: Listing 16.2.7.1

N= Number of subjects in SAS treatment arm, percentages are based on N.

The total number of TEAEs counts all treatment-emergent AEs for subjects. At each level of subject summarization, a subject is counted once for the event with the closest relationship if the subject reported one or more events.

If the relationship of an adverse event is missing, the AE is reported as "Related".

Adverse Events were coded using MedDRA, Version 21.0.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Table 14.3.1. 7 Summary of Treatment-Emergent Serious Adverse Events (Safety Analysis Set)

Source: Listing 16.2.7.5

Repeat table 14.3.1.2 for treatment-emergent serious adverse events

Table 14.3.1. 8 Summary of Treatment- Emergent Related Serious Adverse Events (Safety Analysis Set)

Source: Listing 16.2.7.5

Repeat table 14.3.1.2 for treatment-related emergent serious adverse events

Table 14.3.1.9 Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Analysis Set)

Source: Listing 16.2.7.5

Repeat table 14.3.1.5 for treatment-related emergent serious adverse events

Table 14.3.1. 10 Summary of Treatment-Related Emergent Adverse Events (TEAE) Leading to Discontinuation of the Study (Safety Analysis Set)

Source: Listing 16.2.7.4

Repeat table 14.3.1.2 for treatment-related emergent adverse events leading to discontinuation of the study

Table 14.3.1. 11 Summary of Treatment-Emergent Adverse Events with frequency >= 1% (Safety Analysis Set)

Source: Listing 16.2.7.1

Repeat table 14.3.1.2 for Treatment-Emergent Adverse Events with frequency >= 1%

Table 14.3.1. 12 Summary of Treatment-Emergent Adverse Events with frequency >= 2% (Safety Analysis Set)

Source: Listing 16.2.7.1

Repeat table 14.3.1.2 for Treatment-Emergent Adverse Events with frequency >= 2%

Table 14.3.1. 13 Summary of Treatment-Emergent Adverse Events with frequency >= 3% (Safety Analysis Set)

Source: Listing 16.2.7.1

Repeat table 14.3.1.2 for Treatment-Emergent Adverse Events with frequency >= 3%

Table 14.3.1. 14 Summary of Treatment-Emergent Adverse Events with frequency higher in GSP 301 NS group than in Placebo NS group (Safety Analysis Set)

Source: Listing 16.2.7.1, 16.2.7.2, 16.2.7.3

Repeat table 14.3.1.2 for Treatment-Emergent Adverse Events with frequency higher in GSP 301 NS group than in Placebo NS group

Programming note: for table 14.3.1.11, 14.3.1.12, 14.3.1.13 and 14.3.1.14, frequency for each event is determined by No of subjects that has that event divided by number of subject in the treatment group.

Table 14.3.1. 15 Overall Summary of Adverse Events during Placebo Run-in Period (Run-in Set)

Source: Listing 16.2.7.2

Repeat table 14.3,1,1 for adverse events that occurred in the placebo run-in period, overall column only

Table 14.3.1. 16 Overall Summary of Adverse Events Pre-run-in (All Subjects)

Source: Listing 16.2.7.3

Repeat table 14.3.1.1 for adverse events that occurred in the Pre-run-in Period, overall column only

Table 14.3.2.1.1 Summary of Vital Signs (Safety Analysis Set)

Parameter: Systolic Blood Pressure (mmHg)

| | oo NS | | 01 NS |
|---|---|---|---|
| (N= | xxx) | (N=xxx) | |
| | Change from | | Change from |
| Actual Value | Baseline[a] | Actual Value | Baseline[a] |
| xx (xx) | | xx (xx) | |
| xx.x (xx.xx) | | xx.x (xx.xx) | |
| xx.x | | XX.X | |
| XX, XX | | XX, XX | |
| xx (xx) | | xx (xx) | |
| xx.x (xx.xx) | | xx.x (xx.xx) | |
| xx.x | | xx.x | |
| XX, XX | | XX, XX | |
| xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| xx.x | xx.x | XX.X = | xx.x |
| xx, xx | xx, xx | xx, xx | XX, XX |
| | xx.x (xx.xx) xx.x xx, xx xx (xx) xx.x (xx.xx) xx.x (xx.xx) xx.x xx, xx xx (xx) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) | Actual Value Baseline[a] xx (xx) xx.x (xx.xx) xx.x xx.x xx (xx) xx.x (xx.xx) xx.x xx.x xx (xx) xx (xx) xx (xx) xx (xx) xx (xx) xx (xx) xx.x (xx.xx) xx.x (xx.xx) xx.x xx.x xx.x xx.x xx.x xx.x | Actual Value Baseline[a] Actual Value xx (xx) xx (xx) xx.x (xx.xx) xx.x (xx.xx) xx.x xx.x xx (xx) xx (xx) xx (xx) xx (xx) xx.x (xx.xx) xx.x (xx.xx) xx.x xx.x xx (xx) xx (xx) xx (xx) xx (xx) xx (xx) xx (xx) xx.x (xx.xx) xx.x (xx.xx) xx.x xx.x xx.x xx.x xx.x xx.x |

Source: Listing 16.2.8.5

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the SAS treatment group; n= number of subjects with data available, percentages are based on N.

Baseline is defined as the value collected at Randomization Visit 2.

[a] Change from baseline: post-baseline value – baseline value. For the change from baseline, only subjects with a value at both baseline visit final/discontinuation visit are included.

Program: xxxx.sas Executed: DDMMMYYYYY HH:MM

Glenmark Specialty S.A. Statistical Analysis Plan Study Number - GSP 301-305

December 06, 2018

Programming Note: Repeat table for all VS parameters: diastolic blood pressure (mmHg), pulse rate (BEATS/MIN), height (cm) and weight (kg). Note that height and weight are only collected at baseline and Day 15/Early Termination.

Table 14.3.2.1.2 Summary of Potentially Clinically Significant Vital Signs (Safety Analysis Set)

Parameter: Systolic Blood Pressure (mmHg)

| | | | | Number (9 | %) of subjects | |
|---|---|---|---|---|---|---|
| Treatment Group | Visit | n | n Normal | Abnormal | Abnormal, NCS | Abnormal, CS |
| Placebo NS (N=xxx) | Screening | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 8 | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| GSP 301 NS (N=xxx) | Screening | xx | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 8 | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.8.5

N= Number of subjects in SAS treatment arm; n= Number of subjects that has test for each visit; percentages are based on n.

Baseline is defined as the value collected at Randomization Visit 2.

CS = Clinically Significant; NCS = Not clinically significant

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Vital Sign parameters Systolic blood pressure (mmHg), diastolic blood pressure (mmHg) and pulse rate (BEATS/MIN) will be displayed.

Table 14.3.2.2.1 Summary of Physical Examination (Safety Analysis Set)

General Appearance

| | | | Number (%) of subjects | | | |
|---|---|---|---|---|---|---|
| Treatment Group | Visit | n | Normal | Abnormal | Abnormal, NCS | Abnormal, CS |
| Placebo NS (N=xxx) | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| GSP 301 NS (N=xxx) | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.8.2

N= Number of subjects in SAS treatment arm; n= Number of subjects that has test for each visit; percentages are based on n.

Baseline is defined as the value collected at Screening Visit 1.

CS = Clinically Significant; NCS = Not clinically significant

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat table for all PEs: Neck, head and eyes, cardiovascular system, respiratory system, Musculoskeletal System, Skin, Gastrointestinal System, Genitourinary System, Neurological Examination

Table 14.3.2.3.1 Summary of Focused ENT Examination (Safety Analysis Set)

ENT Examination: Nasal Irritation [a]

| | | Number (%) of subjects | |
|-----------|----------|------------------------|------------|
| Visit | Result | Placebo NS | GSP 301 NS |
| | | (N=xxx) | (N=xxx) |
| Screening | None | xxx (xx.x) | xxx (xx.x) |
| | Grade 1A | xxx (xx.x) | xxx (xx.x) |
| | Grade 1B | xxx (xx.x) | xxx (xx.x) |
| | Grade 2 | xxx (xx.x) | xxx (xx.x) |
| | Grade 3 | xxx (xx.x) | xxx (xx.x) |
| | Grade 4 | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.8.3

N= Number of subjects in SAS treatment arm; percentages are based on N.

Baseline is defined as the value collected at Randomization Visit 2.

[a] Grade 1A and Grade 1B =Mild; Grade 2=Moderate; Grade 3 and Grade 4=Severe

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat table for all ENT examinations follow the value from CRF: Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal Erythema, Crusting of Mucosa, Throat Irritation, Candidiasis and Post Nasal Drip

Table 14.3.2.3.2 Summary of Potentially Clinical Significant Focused ENT Examination (Safety Analysis Set)

ENT Examination: Nasal Irritation

| | Number (%) of subjects | | | | | |
|---|---|---|---|---|---|---|
| Treatment Group | Visit | n | Normal | Abnormal | Abnormal, NCS | Abnormal, CS |
| Placebo NS (N=xxx) | Screening | xx | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 8 | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| GSP 301 NS (N=xxx) | Screening | xx | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 8 | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.8.3

N= Number of subjects in SAS treatment arm; n= Number of subjects that has test for each visit; percentages are based on N.

Baseline is defined as the value collected at Randomization Visit 2.

CS = Clinically Significant; NCS = Not clinically significant

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Repeat table for Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal Erythema, Crusting of Mucosa, Throat Irritation, Candidiasis and Post Nasal Drip

Table 14.3.2.4.1 Summary of Potentially Clinical Significant Eye Examination (Safety Analysis Set)

| | | | Number (%) of subjects | | | |
|---|---|---|---|---|---|---|
| Treatment Group | Visit | n | Normal | Abnormal | Abnormal, NCS | Abnormal, CS |
| Placebo NS (N=xxx) | Screening | xx | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 8 | xx | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| GSP 301 NS (N=xxx) | Screening | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Baseline | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 8 | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Day 15/Early Termination | XX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.8.4

N= Number of subjects in SAS treatment arm; n= Number of subjects that has test for each visit; percentages are based on N

Baseline is defined as the value collected at Randomization Visit 2.

CS = Clinically Significant; NCS = Not clinically significant

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Table 14.3.2.5.1 Summary of Extent of Exposure during the Randomized Treatment Period (Safety Analysis Set)

| | Statistics | Placebo NS<br>(N=xxx) | GSP 301 NS<br>(N=xxx) |
|---|---|---|---|
| Number of Subjects Exposed to Study Treatment n ( | %) | xx (xx.x) | xx (xx.x) |
| Number of Days on Randomized Treatment | n (%) | xx (xx.x) | xx (xx.x) |
| • | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x |
| | Min, Max | xx,xx | xx,xx |
| Number of Days in the Study [a] | n (%) | xx (xx.x) | xx (xx.x) |
| 7 1 1 | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x |
| | Min, Max | xx,xx | xx,xx |
| Randomized Treatment Compliance | < 75% | xxx (xx.x) | xxx (xx.x) |
| * | >= 75% - <= 100% | xxx (xx.x) | xxx (xx.x) |
| | > 100% - <=125% | xxx (xx.x) | xxx (xx.x) |
| | > 125% | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.5.3

SD = Standard Deviation; Max=maximum; Min=minimum; N= number of subjects in the SAS treatment group; n= number of subjects with data available; percentages are based on N.

[a] Number of days on study = End of Study Date - Enrollment Date (Screening Visit) +1

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Listing 16.2.1.1 Listing of Eligibility

| Subject Number | Age(yrs)/<br>Sex/Race | Met all criteria for enrollment? | Inclusion<br>Criteria Not Met | Exclusion<br>Criteria Not Met | Met all criteria for randomi-<br>zation? | Rand Criteria<br>Not Met | Randomization<br>Number |
|---|---|---|---|---|---|---|---|
| 305-000-0001<br>xxx-xxx | 30/F/W<br>xx/x/xx | Yes<br>No | IN01, IN21 | EX02 | | | |
| xxx-xxx-xxx | xx/x/xx | Yes | | | No | RC01 | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Listing 16.2.1.2 Listing of Discontinued Subjects (All Subjects)

| Subject Number | Age(yrs)/<br>Sex/Race | Date of Last Dose<br>Taken (Study Day) | Date of Early Termination/<br>Withdrawal (Study Day) | Reason for Early termination/ Withdrawa |
|---|---|---|---|---|
| 305-000-0001<br>xxx-xxx-xxx | 30/F/W<br>xx/x/xx | dd-mm-yyyy(day)<br>dd-mm-yyyy(day) | dd-mm-yyyy(day)<br>dd-mm-yyyy(day) | Screen Failure<br>Adverse Event |
| xxx-xxx-xxx | xx/x/xx | dd-mm-yyyy(day) | dd-mm-yyyy(day) | XXXXXXXXXXX |
| XXX-XXX-XXX | xx/x/xx | dd-mm-yyyy(day) | dd-mm-yyyy(day) | xxxxxxxxxxx |
| xxx-xxx-xxx | xx/x/xx | dd-mm-yyyy(day) | dd-mm-yyyy(day) | XXXXXXXXXXX |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Programming Note: Continue with treatment group GSP 301 NS.

Page X of Y

Listing 16.2.2.1 Listing of Protocol Deviations (All Subjects)

| Subject Number | Age(yrs)/<br>Sex/Race | Date of Collection<br>(Study Day) | Period | Protocol deviation term | Major [a] |
|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | dd-mm-yyyy(day)<br>dd-mm-yyyy(day) | Treatment<br>Run-In | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes<br>No |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

[a] Subject with major protocol deviation will be exclude from per protocol set.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.3.1 Listing of Subjects Excluded from the Full Analysis Set (Safety Analysis Set)

| Subject Number | Age(yrs)/Sex/Race | Reason for Exclusion |
|---|---|---|
| 305-000-0001 | 30/F/W | Did not have any post-evaluation treatment |
| 305-000-0002 | XX/X/X | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native

Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.3.2 Listing of Subjects Excluded from the Per Protocol Set (Safety Analysis Set)

Treatment Group: Placebo NS

| Subject Number | Age(yrs)/Sex/Race | Reason for Exclusion |
|----------------|-------------------|---------------------------|
| 305-000-0001 | 30/F/W | Did not receive treatment |
| 305-000-0002 | XX/X/X | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYYY HH:MM

Page X of Y

Listing 16.2.4.1 Listing of Demographics (Safety Analysis Set)

| Subject Number | Randomization number | Age | Sex | Race | Ethnicity | Height (cm) | Weight<br>(kg) | BMI<br>(kg/m2) |
|---|---|---|---|---|---|---|---|---|
| 305-000-0001<br>xxx-xxx-xxx | xxxxx | xx | Male<br>Female | Black/ African American<br>White | Not Hispanic or Latino<br>Not Hispanic or Latino | xx.x | xx.x | xx.x |
| <br>XXX-XXX-XXX | | | | | | | | |
| <br>XXX-XXX-XXX | | | | | | | | |
| <br>XXX-XXX-XXX | | | | | | | | |
| 185 | | | | | | | | |

Program: xxxx.sas Executed: DDMMMYYYYY HH:MM

Programming Note: Continue with treatment group GSP 301 NS.

Page X of Y

Listing 16.2.4.2 Listing of Medical History (Safety Analysis Set)

Treatment Group: Placebo NS

| Subject Number | Age(yrs)/<br>Sex/Race | System organ class/ MedDRA preferred term | Description of condition | Start Date/ End<br>Date | Start Day/ End<br>Day | Ongoing at Time of Visit (Screening) |
|---|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXXXX | dd-mm-yyyy /<br>dd-mm-yyyy | xx/xx | No |
| xxx-xxx-xxx | XX/X/X | | | dd-mm-yyyy / | xx/ | Yes |
| XXX-XXX-XXX | | | | | | |
| <br>XXX-XXX-XXX | | | | | | |
| <br>xxx-xxx-xxx | | | | | | |
| 9690 | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Medical History terms were coded using MedDRA, Version 21.0.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Programming Note: Continue with treatment group GSP 301 NS.

Page X of Y

Listing 16.2.4.3 Listing of Prior and Concomitant Medications (Safety Analysis Set)

| Subject<br>Number | Age<br>(yrs)/<br>Sex/<br>Race | Drug Class/<br>Preferred Term/<br>Medication<br>Reported | Flag | Start Date<br>(Day)/<br>Stop Date<br>(Day) | Ongoing | During<br>Run-in<br>Period | During<br>Randomized<br>Treatment<br>Period | Start after Last Study treatment [a] | Dose(Unit)/<br>Route/<br>Freq | Indication |
|---|---|---|---|---|---|---|---|---|---|---|
| 305-000-<br>0001 | 30/<br>F/<br>W | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | P/C | dd-mm-<br>yyyy(day)<br>/<br>dd-mm-<br>yyyy(day) | No | Y/N | Y/N | Y/N | xxx (xx)/<br>Xxx<br>xx | XXXX |
| 30.6 | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | P/C | dd-mm-<br>yyyy(day)<br>/ | Yes | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | | | |
| xxx-xxx-xxx | | XX | | | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Flag: P=Prior medication, C=Concomitant medication; Freq=Frequency

Prior and concomitant medications were coded with the WHO Drug dictionary dated September 2017. Prior medications are medication ended before first randomized treatment. Concomitant medications are medication that are ongoing or ended after first randomized treatment.

Prior medication Day = presented date - first dose date + 1

[a] Start after last randomized treatment.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Sort by Treatment, Subject ID, Start Date/Time, and alphabetically by Drug Class, Preferred Term, and Medication Reported.

December 06, 2018

Listing 16.2.4.4 Listing of Skin Prick Test/Allergy Testing (Safety Analysis Set)

Treatment Group: Placebo NS

| Subject Number | Age(yrs)/<br>Sex/Race | Visit/Test Date (Day) | Object of<br>Observation | Skin Response<br>Test Name | Result (Unit) | Was Allergy testing performed for this visit or within past 12 months? |
|---|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | Screening/dd-mm-yyyy (Day) | Grass | Positive Control | xx.xx (xx) | Yes |

.

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Allergen Testing was performed at Screening Visit (Visit 1) or within the past 12 months

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.4.5 Listing of Pollen Counts and Rainfall by Site (Safety Analysis Set)

| Site name | Collection Date | Type of Allergen | Sub-Category of Type of<br>Allergen | Pollen Count | Did it rain today? | Amount of<br>Rain |
|---|---|---|---|---|---|---|
| 401-XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | dd-mm-yyyy<br>dd-mm-yyyy | Weed<br>Grass | XXXXXXXXX<br>XXXXXXXXX | xxx<br>xxx | Yes<br>No | xx.x |
| 402-XXXXXXXXXXXXXXXXXXXXXXX | dd-mm-yyyy | XXXX<br>XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Listing 16.2.4.6 Listing of Subject Visits (Safety Analysis Set)

| Subject Number | Age(yrs)/<br>Sex/Race | Informed<br>Consent | Screening (Visit 1) | Randomization<br>(Visit 2) | Treatment (Visit 3) | Final/<br>Discontinuation<br>(Visit 4) |
|---|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | dd-mm-yyyy | dd-mm-yyyy | dd-mm-yyyy | dd-mm-yyyy | dd-mm-yyyy |
| xxx-xxx-xxx | xx/x/x | dd-mm-yyyy | dd-mm-yyyy | dd-mm-yyyy | dd-mm-yyyy | dd-mm-yyyy |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.5.1 Listing of Drug Accountability (Safety Analysis Set)

| | | | | | Dispensed | | Return | ed |
|---|---|---|---|---|---|---|---|---|
| | Age(yrs)/ | Date/time of first | T74 1. 3.T | Kit | D : | No. of | D / | No. of |
| Subject Number | Sex/Race | study treatment | Visit Name | Number | Date | bottles | Date | bottles |
| 305-000-0001 | 30/F/W | dd-mm-yyyy(hh:mm) | Screening | xxxxx | dd-mm- | XX | | |
| | | | Randomization | xxxxx | yyyy<br>dd-mm- | xx | dd-mm-yyyy | XX |
| | | | Treatment | xxxxx | уууу<br>dd-mm- | xx | dd-mm-yyyy | XX |
| | | | Final/Discontinuation | ı | уууу | | dd-mm-yyyy | XX |
| XXX-XXX-XXX | | | | | | | | |
| <br>xxx-xxx-xxx | | | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Programming Note: Continue with treatment group GSP 301 NS.

Page X of Y

XXX-XXX-XXX

Listing 16.2.5.2 Listing of Treatment and Dairy Compliance (Safety Analysis Set)

| | | Date/time of first study treatment | | Treatment Co | ompliance | Diary Con | npliance |
|---|---|---|---|---|---|---|---|
| Subject Number | Age(yrs)/<br>Sex/Race | | Visit Name | Subject missed any dose | Number of<br>doses<br>missed | Subject<br>missed any<br>entry | Number<br>of entries<br>missed |
| 305-000-0001 30/F/W | 30/F/W | dd-mm-<br>yyyy(hh:mm) | Treatment | No | | No | |
| | | , | Final/Discontinuation | Yes | 1 | Yes | 2 |
| XXX-XXX-XXX | | | | | | | |
| XXX-XXX-XXX | | | | | | | |
| <br>xxx-xxx-xxx | | | | | | | |
| 225 | | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.5.3 Listing of Extent of Exposure (Safety Analysis Set)

| | | | Treatment | | | Study | |
|---|---|---|---|---|---|---|---|
| Subject Number | Age(yrs)/<br>Sex/Race | First dose Date<br>(Day) / time | Last dose Date<br>(Day) / time | Exposure (days) | Informed<br>Consent date<br>(day) | Completion /<br>discontinuation date<br>(day) | Days in the<br>Study |
| 305-000-0001 | 30/F/W | dd-mm-yyyy(xx) /<br>hh: mm | dd-mm-yyyy(xx) /<br>hh: mm | xx | dd-mm-yyyy(xx) | dd-mm-yyyy(xx) | XX |
| XXX-XXX-XXX | | | | | | | |
| XXX-XXX-XXX | | | | | | | |
| 440 | | | | | | | |
| XXX-XXX-XXX | | | | | | | |
| XXX-XXX-XXX | | | | | | | |
| **** | | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.6.1 Listing of AM and PM Allergic Rhinitis Symptom Evaluation (Reflective Nasal Symptom Scores) (Safety Analysis Set)

| Subject Number | Age(yrs)/<br>Sex/Race | Day | Date | AM/ PM | Dosing<br>Time | Assessment<br>Time | Rhinorrhea | Nasal<br>Congestion | Nasal<br>Itching | Sneezing | rTNSS |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 305-000-0001 | | -7 | dd-mm-yyyy | AM | hh:mm | hh:mm | 0 | 1 | 0 | 0 | 1 |
| | 30/F/W | -6 | dd-mm-yyyy | PM<br>AM | hh:mm | hh:mm | 1 | 1 | 0 | 0 | 2 |
| | | | da-mm-yyyy | PM | | | | | | | |
| | | 14 | dd-mm-yyyy | XX | | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

rTNSS = sum of four reflective nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.6.2 Listing of AM and PM Allergic Rhinitis Symptom Evaluation (Instantaneous Nasal Symptom Scores) (Safety Analysis Set)

| Subject Number | Age(yrs)/<br>Sex/Race | Day | Date | AM/ PM | Dosing<br>Time | Assessment<br>Time | Rhinorrhea | Nasal<br>Congestion | Nasal<br>Itching | Sneezing | iTNSS |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | -7 | dd-mm-yyyy | AM | hh:mm | hh:mm | 0 | 1 | 0 | 0 | 1 |
| | | -6 | dd-mm-yyyy | PM<br>AM<br>PM | hh:mm | hh:mm | 1 | 1 | Ü | U | 2 |
| | | 14 | dd-mm-yyyy | XX | | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native

Hawaiian or Other Pacific Islander, O=Other

iTNSS = sum of four instantaneous nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.6.3 Listing of Subject-reported AM, PM and average AM and PM rTNSS (Safety Analysis Set)

| Subject Number | | | Average AM and PM rTNSS | | | AM rTNSS | | | PM rTNSS | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Age(yrs)/<br>Sex/Race | Day | Baseline[a] | Result | CFB | Baseline[b] | Result | CFB | Baseline[b] | Result | CFB |
| 305-000-0001 | 30/F/W | 1 | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | XX.X | xx.x | XX.X |
| | | 2 | | XX.X | xx.x | | XX.X | xx.x | | XX.X | XX.X |
| | | 3 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |
| | | 18.400 | | | | | | | | | |
| | | 14 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

rTNSS = sum of four reflective nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

CFB = change from baseline.

<sup>[</sup>a] Baseline score of the average AM and PM rTNSS is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization.

<sup>[</sup>b] Baseline score of the AM (PM) rTNSS is derived as the mean of the last 4 consecutive AM (PM) values prior to randomization.

Listing 16.2.6.4 Listing of Subject-reported AM, PM and average AM and PM iTNSS (Safety Analysis Set) Treatment Group: Placebo NS

| Subject Number | | | Average AM and PM iTNSS | | | AN | 1 iTNSS | | PM iTNSS | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Age(yrs)/<br>Sex/Race | Day | Baseline[a] | Result | CFB | Baseline[b] | Result | CFB | Baseline[b] | Result | CFB |
| 305-000-0001 | 30/F/W | 1 | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X |
| | | 2 | | XX.X | xx.x | | XX.X | XX.X | | XX.X | XX.X |
| | | 3 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |
| | | 14 | | xx.x | xx.x | | xx.x | xx.x | | xx.x | xx.x |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

iTNSS = sum of four instantaneous nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing) CFB = change from baseline.

<sup>[</sup>a] Baseline score of the average AM and PM iTNSS is derived as the mean of the last 8 consecutive reading scores.

<sup>[</sup>b] Baseline score of the AM (PM) iTNSS is derived as the mean of the last 4 consecutive AM (PM) values prior to randomization.

Listing 16.2.6.5 Listing of AM and PM Reflective Non-Nasal Symptom Scores (Safety Analysis Set)

| Subject Number | Age(yrs)/<br>Sex/Race | Day | Date | AM/<br>PM | Assessment<br>Time | Itching/<br>Burning<br>Eyes | Tearing/<br>Watering<br>Eyes | Redness<br>of Eyes | Itching<br>of Ears<br>or<br>Palate | rTNNSS | rTOSS |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | -7 | dd-mm-yyyy | AM<br>PM | hh:mm<br>hh:mm | 0 | 1 | 0 | 1 0 | 2 | 1 |
| | | -6<br><br>14 | dd-mm-yyyy<br>dd-mm-yyyy | AM<br>PM<br>XX | 111111111 | 1 | 1 | v | 0 | 2 | 2 |

rTNNSS = sum of four reflective non-nasal symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes, Itching of Ears or Palate) rTOSS = sum of three reflective non-nasal symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes)

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.6.6 Listing of AM and PM Instantaneous Non-Nasal Symptom Scores (Safety Analysis Set)

| Subject Number | Age(yrs)/<br>Sex/Race | Day | Date | AM/<br>PM | Assessment<br>Time | Itching/<br>Burning<br>Eyes | Tearing/<br>Watering<br>Eyes | Redness<br>of Eyes | Itching<br>of Ears<br>or<br>Palate | iTNNSS | iTOSS |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | -7 | dd-mm-yyyy | AM<br>PM | hh:mm<br>hh:mm | 0 | 1 | 0 | 1 | 2 2 | 1 2 |
| | | -6<br><br>14 | dd-mm-yyyy<br>dd-mm-yyyy | AM<br>PM<br>XX | | | | | | | |

iTNNSS = sum of four instantaneous non-nasal symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes, Itching of Ears or Palate) iTOSS = sum of three instantaneous non-nasal symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes)

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y
Listing 16.2.6.7 Listing of Subject-reported AM, PM and average AM and PM rTNNSS (Safety Analysis Set)

| | | | Average AN | I and PM r | TNNSS | AM | rTNNSS | | PM rTNNSS | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Number | Age(yrs)/<br>Sex/Race | | Baseline[a] | Result | CFB | Baseline[b] | Result | CFB | Baseline[b] | Result | CFB |
| 305-000-0001 | 30/F/W | 1 | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | XX.X |
| | | 2 | | XX.X | XX.X | | XX.X | xx.x | | XX.X | XX.X |
| | | 3 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |
| | | 14 | | xx.x | xx.x | | xx.x | XX.X | | xx.x | xx.x |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

rTNNSS = sum of four reflective non-nasal symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes, Itching of Ears or Palate).

CFB = change from baseline.

<sup>[</sup>a] Baseline score of the average AM and PM rTNNSS is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization.

<sup>[</sup>b] Baseline score of the AM (PM) rTNNSS is derived as the mean of the last 4 consecutive AM (PM) values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

Listing 16.2.6.8 Listing of Subject-reported AM, PM and average AM and PM iTNNSS (Safety Analysis Set)

| | | | Average AN | 1 and PM i | TNNSS | AM | iTNNSS | | PM iTNNSS | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Number | Age(yrs)/<br>Sex/Race | _ | Baseline[a] | Result | CFB | Baseline[b] | Result | CFB | Baseline[b] | Result | CFB |
| 305-000-0001 | 30/F/W | 1 | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| | | 2 | | xx.x | XX.X | | xx.x | XX.X | | XX.X | XX.X |
| | | 3 | | XX.X | XX.X | | xx.x | XX.X | | XX.X | XX.X |
| | | 14 | | | | | | | | | |
| | | 14 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |

iTNNSS = sum of four instantaneous non-nasal symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes, Itching of Ears or Palate). CFB = change from baseline.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

<sup>[</sup>a] Baseline score of the average AM and PM iTNNSS is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization.

<sup>[</sup>b] Baseline score of the AM (PM) iTNNSS is derived as the mean of the last 4 consecutive AM (PM) values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

Listing 16.2.6.9 Listing of Subject-reported AM, PM and average AM and PM rTOSS (Safety Analysis Set)

| | | | Average Al | M and PM | rTOSS | AN | 1 rTOSS | | PN | 1 rTOSS | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Number | Age(yrs)/<br>Sex/Race | Day | Baseline[a] | Result | CFB | Baseline[b] | Result | CFB | Baseline[b] | Result | CFB |
| 305-000-0001 | 30/F/W | 1 | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | XX,X | xx.x | xx.x |
| | | 2 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |
| | | 3 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | xx.x |
| | | 8697 | | | | | | | | | |
| | | 14 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

rTOSS = sum of three reflective ocular symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes).

CFB = change from baseline.

<sup>[</sup>a] Baseline score of the average AM and PM rTOSS is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization.

<sup>[</sup>b] Baseline score of the AM (PM) rTOSS is derived as the mean of the last 4 consecutive AM (PM) values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

Listing 16.2.6.10 Listing of Subject-reported AM, PM and average AM and PM iTOSS (Safety Analysis Set)

Treatment Group: Placebo NS

| | | | Average Al | M and PM | iTOSS | AM | 1 iTOSS | | PN | 1 iTOSS | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Number | Age(yrs)/<br>Sex/Race | | Baseline[a] | Result | CFB | Baseline[b] | Result | CFB | Baseline[b] | Result | CFB |
| 305-000-0001 | 30/F/W | 1 | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | XX.X |
| | | 2 | | xx.x | XX.X | | XX.X | XX.X | | XX.X | XX.X |
| | | 3 | | XX.X | XX.X | | XX.X | XX.X | | XX.X | XX.X |
| | | 14 | | xx.x | xx.x | | xx.x | xx.x | | xx.x | XX.X |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

iTOSS = sum of three reflective ocular symptom scores (Itching/Burning Eyes, Tearing/Watering Eyes, Redness of Eyes).

CFB = change from baseline.

<sup>[</sup>a] Baseline score of the average AM and PM iTOSS is derived as the mean of the last 8 consecutive reading scores including the AM assessment on the day of randomization.

<sup>[</sup>b] Baseline score of the AM (PM) iTOSS is derived as the mean of the last 4 consecutive AM (PM) values prior to randomization during the last 4 days of the run-in period from the Day -4 PM assessment to the AM assessment on the day of randomization.

Listing 16.2.6.11 Listing of Pediatric Rhinoconjunctivitis Quality of Life (PRQLQ) (Safety Analysis Set)

| Treatment | Group: | Placebo | NS |
|-----------|--------|---------|----|
|-----------|--------|---------|----|

| | | | | | NC | )SE | | - | E. | YE | | | PRACTI | CAL PR | OBLEMS | 5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Age(yrs)/<br>Sex/Race | Visit | Date | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 | Q11 | Q12 | Q20 |
| 305-<br>000-<br>0001 | 30/F/W | Randomization | | | | | | | | | | | | | | |
| 0001 | | Day 15 | | | | | | | | | | | | | | |

| Subject | ubject Age(yrs)/ | | | OTHER SYMPTOMS | | | | | ACTIVITY LIMITATION | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Sex/Race | Visit | Date | Q13 | Q14 | Q15 | Q17 | Q18 | Q19 | Q16 | Q21 | Q22 | Q23 |
| 305-000- | 30/F/W | Randomization | | | | | | | | | | | |
| 0001 | | Day 15 | | | | | | | | | | | |

Baseline is defined as the time point "pre-dosing" at the Randomization Visit (Visit 2). Day 15 includes Visit 4 for all subjects, including those terminating early, regardless of what actual study day this visit occurred on.

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.6.12 Listing of Physician Assessed Nasal Symptom Scores (PNSS) (Safety Analysis Set)

| Subject | Age(yrs)/ | | | Nasal | Nasal | | | Change from |
|---|---|---|---|---|---|---|---|---|
| Number | Sex/Race | Visit | Rhinorrhea | Congestion | Itching | Sneezing | PNSS | Baseline |
| | | Randomization | 0 | 1 | 0 | 0 | 1 | |
| 305-000-0001 | 30/F/W | Day 15 | 1 | 1 | 0 | 0 | 2 | 1 |

Baseline is defined as the time point "pre-dosing" at the Randomization Visit (Visit 2)

PNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

149

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.7.1 Listing of Treatment Emergent Adverse Events by Treatment During Randomized Treatment Period (Safety Analysis Set)

| Treatment Group: | Placebo NS | | | | | |
|---|---|---|---|---|---|---|
| | | System Organ Class/ | Start Date<br>(Day)/<br>End Date | Severity/<br>Relationship/ | Outcome / | Cause |
| Subject<br>Number | Age(yrs)/<br>Sex/Race | Preferred Term [c]/ Verbatim Term | (Day)/<br>Duration | Action Taken with IP | Additional<br>Treatment Given | Discontinuation/<br>Serious AE |
| 305-000-0001 | 30/F/W | NERVOUS SYSTEM<br>DISORDERS/ HEADACHE/<br>HEADACHE* | dd-mm-yyyy<br>(Day)/<br>dd-mm-yyyy<br>(Day)/ | Mild/<br>Not Related/<br>None | Recovered or Resolved<br>with Sequelae/<br>No | No/ No |
| | | | XX | | | |

<sup>\*=</sup>Treatment-emergent AE

Day = The presented date – First dose date + 1

Duration (Days = Stop date – Start date + 1)

Adverse Events were coded using MedDRA, Version 21.0

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Programming Note: Continue with treatment group GSP 301 NS.

Listing 16.2.7.2 Listing of Adverse Events During Placebo Run-in Period (Run-in Set)

Repeat Listing 16.2.7.1 for Placebo run-in period for overall. Remove "Treatment group:xxx" on top of the table.

Listing 16.2.7.3 Listing of Adverse Events During Pre-run-in Period (All Subjects)
Repeat Listing 16.2.7.1 for Pre-run-in Period for overall. Remove "Treatment group:xxx" on top of the table.

Listing 16.2.7.4 Listing of Adverse Events Leading to Withdrawal (All Subjects) Repeat Listing 16.2.7.1 for adverse events Leading to Withdrawal

Listing 16.2.7.5 Listing of Serious Adverse Event During Randomized Treatment Period (Safety Analysis Set) Repeat Listing 16.2.7.1 for Serious Adverse events

Listing 16.2.7.6 Listing of Serious Adverse Event During Placebo Run-in Period (Run-in Set)

Repeat Listing 16.2.7.1 for Serious Adverse events during Placebo run-in period for overall. Remove "Treatment group:xxx" on top of the table.

Listing 16.2.7.7 Listing of Serious Adverse Event During Pre-run-in Period (All Subjects)

Repeat Listing 16.2.7.1 for Serious Adverse events during Pre-run-in Period for overall. Remove "Treatment group:xxx" on top of the table.

Glenmark Specialty S.A. Statistical Analysis Plan Study Number - GSP 301-305

December 06, 2018

## Listing 16.2.7.8 Listing of Death (All Subjects)

Treatment Group: Placebo NS

| Subject<br>Number | Age(yrs)/<br>Sex/Race | Date of Death (Day) | Cause of Death |
|---|---|---|---|
| 305-000-0001 | 30/F/W | dd-mm-yyyy (Day) | xxxx |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.8.1 Listing of Pregnancy Test Results (Safety Analysis Set)

| Subject Number | Age(yrs)/<br>Sex/Race | Visit | Was Urine Pregnancy Test Performed? | Date (Day) | Result | Reason Not done |
|---|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | Screening | | dd-mm-yyyy | | |
| | | | Yes | (Day) | Negative | |
| | | Randomization | No | | | XXXXXXXXXXXXXXXXXXXXXXX |
| | | Day 15 | | dd-mm-yyyy | | |
| | | | Yes | (Day) | Negative | |

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Programming Note: Continue with treatment group GSP 301 NS.

153

Listing 16.2.8.2 Listing of Physical Examination (Safety Analysis Set)

| Treatment | Group: | Placebo NS |
|----------------|---------|---------------|
| I I Catillolli | OI OUD. | I Idocoo I ID |

| | Age(yrs)/ | Visit/ | | | Clinical | Abnormality |
|---|---|---|---|---|---|---|
| Subject Number | Sex/Race | Exam Date(Day) | Assessment | Result | Significance | Comment(s) |
| 305-000-0001 | 30/F/W | Screening/<br>dd-mm-yyyy(day) | General Appearance | Abnormal | NCS | XXXXXXXX |
| | | | Neck | Normal | | |
| | | | Head and Eyes | Normal | | |
| | | | Cardiovascular System | Normal | | |
| | | | Respiratory System | Normal | | |
| | | | Musculoskeletal System | Normal | | |
| | | | Skin | Normal | | |
| | | | Gastrointestinal System | Normal | | |
| | | | Genitourinary System | Normal | | |
| | | | Neurological Examination | Normal | | |
| | | | Other | Normal | | |
| | | <repeat 15="" day="" for=""></repeat> | | | | |
| xxx-xxx-xxx | | | | | | |

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Clinical Significance: CS = Clinically Significant; NCS = Not Clinically Significant

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Programming Note: Continue with treatment group GSP 301 NS.

Listing 16.2.8.3 Listing of Focused ENT Examination (Safety Analysis Set)

| Treatment | Group: | Place | bo NS |
|-----------|--------|-------|-------|

| Subject Number | Age(yrs)/<br>Sex/Race | Visit/Exam Date<br>(Day) | Evaluation | Result | Clinical<br>Significance |
|---|---|---|---|---|---|
| 305-000-0001 | 30/F/W | Screening/<br>dd-mm-yyyy(day) | Nasal Irritation | Grade1B = Superficial mucosal erosion | NCS |
| | | | Epistaxis | Mild | NCS |
| | | | Mucosal Edema | None | NCS |
| | | | Nasal Discharge | Mild | NCS |
| | | | Mucosal Erythema | Mild | NCS |
| | | | Crusting of Mucosa | Mild | NCS |
| | | | Throat Irritation | Present | NCS |
| | | | Candidiasis | Absent | NCS |
| | | | Post Nasal Drip | Absent | NCS |
| | | <repeat for<br="">Randomization<br/>Day 8<br/>Day 15&gt;</repeat> | | | |
| ···<br>xxx-xxx-xxx | | | | | |

AAA-AAA-AAA

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native

Hawaiian or Other Pacific Islander, O=Other

Clinical Significance: CS = Clinically Significant; NCS = Not Clinically Significant

Program: xxxx.sas Executed: DDMMMYYYY HH:MM

Page X of Y

Listing 16.2.8.4 Listing of Eye Examination (Safety Analysis Set)

| | Age(yrs)/ | Visit/Exam | | | Description | |
|---|---|---|---|---|---|---|
| Subject Number | Sex/Race | Date (Day) | Side of Eye | Result | of Abnormality | Clinical Significance |
| 305-000-0001 | 30/F/W | Screening/<br>dd-mm-<br>yyyy(day)<br>< Repeat for<br>Randomization<br>Day 8<br>Day 15> | Left | Normal | xxx | NCS |
| *** | | | | | | |

XXX-XXX-XXX

Sex: M=Male, F=Female; Race: W=White, BL=Black or African American, AS=Asian, AI=American Indian or Alaska Native, ML=Multiple, PI=Native Hawaiian or Other Pacific Islander, O=Other

Clinical Significance: CS = Clinically Significant; NCS = Not Clinically Significant

Program: xxxx.sas Executed: DDMMMYYYYY HH:MM

Programming Note: Continue with treatment group GSP 301 NS.

Listing 16.2.8.5 Listing of Vital Signs (Safety Analysis Set)

| Subject Number | Visit | Collection Date (Day) | Vital Sign Parameter | Position | Result | Units | Flag/ Clinical<br>Significance |
|---|---|---|---|---|---|---|---|
| 305-000-0001 | Screening | dd-mm-yyyy (Day) | Systolic Blood Pressure Diastolic Blood Pressure Pulse Rate Height Weight | Sitting<br>Sitting | xx.x<br>xx.x | mmHg<br>mmHg<br>BPM<br>cm<br>kg | Normal<br>Ab; NCS<br>Normal |
| | Randomization | dd-mm-yyyy (Day) | Systolic Blood Pressure Diastolic Blood Pressure Pulse Rate | Sitting<br>Sitting | xx.x<br>xx.x | mmHg<br>mmHg<br>BPM | Normal<br>Normal<br>Normal |
| | Day 8<br>Day 15 | | | | | | |

Flag: Ab;NCS=Abnormal;Not Clinically Significant, Ab;CS=Abnormal;Clinically Significant

Program: xxxx.sas Executed: DDMMMYYYY HH:MM